# **CLINICAL PROTOCOL**

A Phase II, Placebo-Controlled, Randomized, Double-Blind Study to Assess the Safety, Tolerability and Efficacy of terpenes-enriched CBD-predominant cannabis oil, Administered to Pediatric Subjects with Autism Spectrum Disorder (ASD)

**Protocol Number:** 0336-24-SZMC

Investigational Product: Terpenes-enriched cannabis oil T1/C28

**Protocol Version:** September 1, 2025, Version 3.0

ClinicalTrials.gov Identifier: NCT07199218

| Prepared by: | Title | Date | Signature |
|--------------|------------------------|------------|-----------|
| Adi Aran, MD | Principal Investigator | 01/09/2025 | |

# **Revision History – After recruitment of first patient**

| Version | Author | Date | Description |
|---------|--------|------|-------------|

# **Short Synopsis**

| Title | A Phase 2, Placebo-Controlled, Randomized, Double-Blind Study to Assess the |
|---|---|
| | Safety, Tolerability and Efficacy of terpenes-enriched cannabis oil T1/C28, |
| | Administered to Pediatric Subjects with Autism Spectrum Disorder (ASD) |
| Short Title | A placebo-controlled trial of terpenes-enriched CBD-predominant cannabis oil in children with ASD |
| Running Head | Terpenes-enriched CBD oil in ASD |
| Protocol Number | 0336-24-SZMC |
| Study Center | Shaare Zedek Medical Center, Jerusalem, Israel |
| CinicalTrials.gov Identifier | NCT07199218 |
| - Registration Date | September 29, 2025 |
| <b>Ethic Approval Date</b> | May 25, 2025 |
| Trial Commencement | TBD |
| Planned Number of Participants | 78 |
| Study duration per participant | Placebo-controlled phase: 8 weeks; After completing the first 8-week period, participants who received placebo will receive terpenes-enriched CBD, and participants who received the study drug will continue with the same treatment for another 8 weeks. |
| <b>Study Intervention</b> | Cannabidiol (CBD; 7.2mg/kg/d); Tetrahydrocannabinol (THC; 0.257mg/kg/d); and Terpenes (0.5mg/kg/d). Study intervention will be administered separately <b>as an add-on</b> to any existing treatment. |
| Primary outcome | ASD-associated behavioral problems, using the Aberrant Behavior Checklist-Irritability Subscale (ABC-I) score - change from baseline to week 8. |

# Contents

| 1. | Title page | 1 |
|---|---|---|
| 2. | Revision history Short synopsis | 2 |
| 3. | Contents | 4 |
| 4. | Abstract | 5 |
| 5. | Introduction | 7 |
| 6. | Hypotheses and Significance | 10 |
| 7. | Study Design | 10 |
| 8. | Subjects | 12 |
| 9. | Procedures | 12 |
| 10. | Outcomes and Measures | 14 |
| 11. | Assessment schedule | 18 |
| 12. | Study Flow Chart | 19 |
| 13. | Statistical Considerations. | 20 |
| 14. | Data Management | 24 |
| 15. | Informed Consent Process, Vulnerable Population and DSMB | 24 |
| 16. | Randomization and blinding | 25 |
| 17. | Study Interventions, Dose Justification and Administration | 26 |
| 18. | Amendments to the protocol & Deviations from the protocol | 27 |
| 19. | Statement Of Compliance, Eearly Termination, and Publication Policy | 28 |
| 20. | Adverse Events | 29 |
| 21. | Appendix 1 – Non-Generic Questionaires | 30 |
| 22. | Appendix 2 – Detailed summary of previous related randomised studies | 39 |
| 23. | Bibliography | 40 |

# A Placebo-Controlled Trial of Terpenes-Enriched, Cannabidiol-Predominant Cannabis Oil in Children with ASD

Background: Autism spectrum disorder (ASD) encompasses a wide range of neurodevelopmental disorders with diverse etiologies and symptoms. Efforts to develop a single pharmacological treatment for the core symptoms of ASD have been unsuccessful. Approved antipsychotic medications for managing associated irritability often result in substantial metabolic side effects. Cannabidiol (CBD), a non-psychoactive cannabinoid, targets multiple neuronal and glial pathways to reduce excitation and inflammation. In contrast, tetrahydrocannabinol (THC), a psychoactive cannabinoid, directly activates the endocannabinoid system, which is impaired in ASD, and decreases social anxiety and hostility. Preliminary trials in children with ASD have demonstrated the efficacy of a CBD-predominant formulation combined with low-dose THC. Preclinical data suggest that efficacy may be further enhanced by enriching cannabinoid compounds with selected terpenes, which activate CB1 and CB2 receptors both directly and by modulating THC interactions at these receptors.

**Objective:** To assess the impact of terpenes-enriched, CBD-predominant, cannabis oil on children with ASD in a randomized, double-blind, placebo-controlled trial.

### Specific aims:

<u>The primary aim</u> is to assess the effect of the study drug compared to placebo on behavioral problems, using the Aberrant Behavior Checklist-Irritability Subscale (ABC-I) score - change from baseline to week 8.

The main secondary aim is to assess the effect of the study drug compared to placebo on core ASD symptoms using the Vineland <sup>TM</sup> Adaptive Behavior Scales (3rd edition, VABS3)-Socialization Domain Score, and the Social Responsiveness Scale 2nd edition (SRS-II) total score - change from baseline to week 8.

Other secondary aims include: (1) To assess the tolerability and safety of the study drug compared to placebo, using detailed questionnaires, physical examination, blood count, and liver enzyme tests. (2) To assess global change in ASD-associated symptoms since baseline using the Clinical Global Impression- Improvement (CGI-I) and the Caregiver Global Impression of Change (CGIC) assessments – at week 8. (3) To assess changes in the quality of life, sleep parameters, and gastrointestinal problems using the Quality of Life in Autism Questionnaire (QOLA) – Parent version, the Children's Sleep Habits Questionnaire (CSHQ) and a modified gastrointestinal sign and symptoms inventory (GISSI) - change from baseline to week 8. (4) To compare the effect of CBD-predominant, cannabis oil (study drug) with terpenes-enriched CBD, using the above assessments - change from baseline to week 8 and week 17.

**Study design:** In this phase 2, randomized, double-blind, placebo-controlled, parallel-group study,78 children with ASD and behavioral problems, will be randomized (in a 1:1 ratio) to receive either placebo or a terpenes-enriched CBD-predominant cannabis oil (CBD 7.2mg/kg/d; THC 0.257mg/kg/d; Total terpenes 0.5mg/kg/d). The treatment will be given as an add-on to any existing treatment, for 8 weeks. The treatment dose will be up-titrated over 8days. After completing the first 8-week period, participants who received placebo will receive terpenes-enriched pure CBD, and participants who received the study drug will continue with the same treatment for another 8 weeks.

Inclusion criteria: A diagnosis of ASD according to the DSM-5 criteria; Age 4-12 years; Bodyweight between 12.5kg and 57.5kg; CGI-Severity score ≥ 4; ABC-I score ≥ 18; and SRS-II total T score > 66.

<u>Exclusion criteria</u>: Seizures or changes in anticonvulsive therapy within the last 16 weeks; Treatment with cannabinoids or any change in the pharmacological or behavioral treatment in the

September 1, 2025, Version 3.0 Confidential and Proprietary

4 weeks prior to randomization; Participants or caregivers are unlikely (in the investigator's opinion) to comply with all trial requirements including blood tests.

**Significance:** Previous studies suggest that CBD-rich cannabis oil (CBD:THC ratio = 20:1) reduces disruptive behavior and improves core symptoms in children with ASD. However, THC use remains controversial. While whole-plant extracts may enhance benefits via the "entourage effect" (synergy of cannabinoids and terpenes), cannabinoid isolates offer precise and consistent dosing. Enriching cannabinoid isolates with selected terpenes preserves the entourage effect and enables reducing THC dosage while ensuring both efficacy and consistency.

# **Introduction**

There is no established pharmacological treatment for the core symptoms of autism spectrum disorder (ASD), persistent deficits in social communication, and repetitive, restrictive patterns of behavior. Risperidone and aripiprazole have been approved by the U.S. Food and Drug Administration (FDA) to treat comorbid irritability² but these medications often cause obesity and metabolic syndrome. Additionally, Up to 80% of children with ASD also have sleep disorders. Cannabinoid therapy with various THC to CBD ratios is being increasingly used to alleviate sleep disorders regardless of cause. However, currently there is insufficient evidence to support this line of treatment.

Cannabinoids, have been assessed before to treat core and comorbid symptoms in children with ASD with mixed results. 10

The partial effects demonstrated in these studies can be attributed to the heterogeneous and multifactorial etiology of ASD which should probably better be addressed with polytherapy. The current study aims to assess the combined impact of cannabidiol (CBD), terpenes and low-dose THC which target multiple key biochemical hubs in antioxidative, anti-inflammatory, and cytoprotective pathways. <sup>10</sup>

We hypothesize that combined treatment with these 3 compounds will lead to significantly higher improvement in disruptive behavior and core autistic symptoms compared with placebo in children with ASD.

The endocannabinoid system is a cell-signaling system composed of the cannabinoid receptors, their endogenous ligands [*endocannabinoids, mainly* anandamide (AEA) and 2-AG], transporters, and enzymes that produce and degrade the endocannabinoids.<sup>11</sup>

Studies in animal models suggest a reduced endocannabinoid tone in ASD. 12-16 Stimulation of the endocannabinoid system 12-17 have improved social deficits in some models. Additionally, children with ASD have lower peripheral endocannabinoid levels. 16,18,19

The main components of the cannabis plant (phytocannabinoids) are Δ9-tetrahydrocannabinol (THC) and cannabidiol (CBD). THC activates the type-1 cannabinoid receptor (CB<sub>1</sub>R) – the main cannabinoid receptor in neurons (Figure 1). THC is psychoactive (causes a 'high' feeling) and can lead to anxiety, addiction, cognitive decline, motivational loss, and psychosis. <sup>20</sup> CBD, on the other hand, is a negative allosteric modulator of the CB<sub>1</sub>R which decreases the effects of CB<sub>1</sub>R agonists such as THC. Nevertheless, CBD can activate the endocannabinoid system by decreasing the reuptake of the endocannabinoids (AEA and 2-AG) and the degradation of AEA (Figure 1). CBD is not psychoactive and has a relatively high toxicity threshold. <sup>20</sup> It also appears to have anxiolytic, antipsychotic, antiepileptic, and neuroprotective properties that may be mediated through receptors such as serotonin 5-HT<sub>1A</sub>, TRPV1, GPR55, GABA<sub>A</sub>, D2, and PPARγ, and by inhibiting adenosine reuptake (Figure 1). <sup>21-25</sup>

Besides its direct effects on multiple receptor targets in neurons, CBD has prominent direct and indirect antioxidant and immunomodulatory effects<sup>26-33</sup> that were extensively studied in microglia<sup>34-37</sup> (Figure 2). Immune system dysregulation has a direct impact on numerous neurodevelopmental processes.<sup>38</sup> In ASD, immune dysregulation includes differential monocyte, macrophage, and microglia responses,<sup>39-44</sup> and abnormal cytokine, and T cell levels.<sup>38,45,46</sup> Additionally, in most of the ASD cases, there are indications of mitochondrial function impairments including lactic acidemia, abnormal lactate: pyruvate ratios, and accumulation of alanine in the plasma and urine indicating defects in oxidative phosphorylation.<sup>47-49</sup> Hence, the immunomodulatory and antioxidative effects of CBD and its effects on the endocannabinoid system and various other receptors could be beneficial in ASD. Previously, we demonstrated in a placebo-controlled trial that a CBD-rich cannabis extract (with a CBD-to-THC ratio of 20:1) can reduce disruptive behaviors associated with ASD and improve core autistic symptoms with acceptable tolerability.<sup>50</sup> However, due to the potential risks of THC,

particularly in children with neuropsychiatric disorders, ongoing and emerging placebo-controlled studies are focusing on the effects of CBD isolates devoid of THC.<sup>51</sup>

Nevertheless, animal studies,<sup>17</sup> preliminary evidence from randomised studies,<sup>10</sup> and our clinical experience suggest that CBD alone has significantly lower efficacy. Recent preliminary clinical and preclinical studies indicate that efficacy might be enhanced by enriching CBD-dominant compounds with specific terpenes. These terpenes can activate CB1 and CB2 receptors directly or modulate THC interactions with these receptors.<sup>52-57</sup>

In the current study, we aimed to evaluate the efficacy, safety, and tolerability of terpeneenriched, CBD-predominant cannabis oil with a CBD-to-THC ratio of 28:1



**Figure 1:** The main cannabinoid receptor in neurons is the Cannabinoid receptor type-1 ( $CB_1R$ ). Activated  $CB_1R$  increases outflow of potassium and decreases inflow of calcium reducing synaptic transmission. THC directly activates the  $CB_1R$ . Specific terpenes directly activate the  $CB_1R$  and increase  $CB_1R$  activation by THC. CBD is a negative allosteric modulator of the  $CB_1R$ . However, CBD can activate the endocannabinoid system by inhibiting the endocannabinoid membrane transporter (EMT) and the degradation of anandamide (AEA) through Fatty acid amide hydrolase (FAAH). This, in turn, increases the levels of the endocannabinoids AEA (a main agonist of  $CB_1R$ ) and 2-Arachidonoylglycerol (2-AG). Other neuronal effects of CBD are mediated through full agonism at 5- $HT_{1A}$  serotonin receptors and TRPVI channel reducing anxiety and pain; Partial agonism at D2 dopamine receptors increasing emotional regulation; A negative allosteric modulation of MOR reducing opioid drug abuse and relapse; and Agonism of the nuclear  $PPAR\gamma$  receptors increasing expression of cytoprotective enzymes. CBD also has direct antioxidative effects.

D2: dopamine receptor 2; ENT: equilibrative nucleotide transporter; 5-H $T_{IA}$ : 5-hydroxytryptamine 1A receptor; GPR55: G protein-coupled receptor 55; MOR:  $\mu$  opioid receptor; PPARy: peroxisome proliferator-activated receptor gamma; ROS, reactive oxygen species; TRPV1: transient receptor potential vanilloid 1.



Figure 2: Molecular targets of CBD in microglia. CBD has anti-inflammatory and antioxidative effects in the microglia which are mostly not related to the cannabinoid receptors. CBD is a full agonist of adenosine  $A_2A$ , and the TRPV1 cell membrane receptors and the nuclear PPARy receptor – all convey anti-inflammatory effects. PPARy is a ubiquitin E3 ligase that leads to proteasomal degradation of the p65 subunit of the proinflammatory transcription factor nuclear factor kappa B (NF- $\kappa$ B). In the nucleus, PPARy reduces the expression of proinflammatory cytokines and increases the expression of anti-inflammatory and anti-oxidative mediators. CBD also has direct antioxidative effects. The main cannabinoid receptor in microglia is Cannabinoid receptor type-2 ( $CB_2R$ ). Expression of  $CB_2R$  is upregulated in reactive microglia. The main effect of the CB<sub>2</sub>R is anti-inflammatory. While initially activating the proinflammatory mediators of the mitogen-activated protein kinase (MAPK) family,  $CB_2R$  prevents further activation of MAPK by powerful triggers such as lipopolysaccharide (LPS). CBD has a weak affinity to the CB<sub>2</sub>R (mostly as an inverse agonist). However, CBD can activate the endocannabinoid system through the CB<sub>2</sub>R by inhibiting the endocannabinoid membrane transporter (EMT) which leads to reuptake inhibition of 2-Arachidonoylglycerol (2-AG) the main agonist of  $CB_2R$ .

ENT: equilibrative nucleotide transporter; GDNF: a glial cell line-derived neurotrophic factor; GPR55: G protein-coupled receptor 55; PPAR $\gamma$ : peroxisome proliferator-activated receptor gamma; ROS, reactive oxygen species; TNF- $\alpha$ , tumor necrosis factor-alpha; TRPV1: transient receptor potential vanilloid I

### **Working hypothesis and expected significance:**

In the proposed study, we will assess the effects of CBD and low-dose THC isolates, enriched with selected terpenes, on alleviating disruptive behavior and core symptoms in children with ASD. Combination therapy is anticipated to achieve higher efficacy compared to monotherapy and is a standard of care in many medical disorders, including cancer and cardiovascular disease. CBD and terpenes are plant-derived compounds with high safety and tolerability, possessing proven anti-inflammatory, antioxidative, and mitochondrial-supportive properties. These compounds have shown promising preliminary efficacy in ASD trials.

THC directly activates the endocannabinoid system, which has been shown to be impaired in ASD. Due to concerns regarding THC safety in children, we will use a lower THC dose in this study (0.27 mg/kg/day) compared to our previous study, where a dose of 0.5 mg/kg/day was used. We hypothesize that this combination of compounds will lead to significantly greater improvements in disruptive behavior and core autistic symptoms compared to placebo. The use of cannabinoid isolates enriched with terpenes, rather than whole-plant extracts (which can vary by batch), will ensure consistency of treatment and allow for a substantial increase in the dose of terpenes, the safest component of the formulation.

Despite the efficacy of atypical antipsychotics (mainly risperidone) in treating behavioral problems in individuals with ASD,<sup>58-60</sup> approximately 40% of patients experience drug-refractory aggression, self-injurious behavior, and severe tantrums.<sup>61</sup> Furthermore, risperidone and other atypical antipsychotics are associated with substantial adverse effects, such as sleepiness and weight gain. Consequently, many patients continue to suffer from disruptive behaviors that significantly impact their daily functioning and place a heavy burden on their caregivers. Even a minor improvement in the severity of ASD core and associated symptoms can have a profound impact on the lives of countless families and reduce public health costs.

### Methods

#### Study design

This is a phase 2, randomized, double-blind, placebo-controlled, parallel-group study, involving 78 children with ASD and behavioral problems, age 4-12 years. Participants who will pass screening will be randomized (in a 1:1 ratio) to receive either placebo or terpenes-enriched CBD rich cannabis oil (CBD: 3.6 mg/kg twice daily, terpenes: 0.25mg/kg twice daily, and THC: 0.128 mg/kg twice daily). The treatment will be given orally as an add-on to any existing treatment, for 8 weeks. The treatment dose will be up-titrated over 8 days.

After completing the first 8-week period, participants who received placebo will receive pure CBD (3.6 mg mg/kg twice daily enriched with terpenes (0.25mg/kg twice daily), and participants who received the study drug will continue with the same treatment for another 8 weeks of the second phase. (Figure 3).

#### First phase

Every 4 days during the titration phase and every 2 weeks thereafter, parents or primary caregivers will rate adverse events and document: any use of medical services, any change in the doses of the study intervention and concomitant medications, any change in the regular diet and intake of food supplements, and any change in the home or school routine or in the behavioral or emotional treatments.

Additionally, at each study visit, physicians will assess physical examination and BMI, and parents or primary caregivers will rate behavioral symptoms on the Aberrant Behavior Checklist-Community (ABC-C) – Irritability subscale (ABC-I) and ASD core symptoms on the Social Responsiveness Scale – second edition (SRS-2).

### Other assessments at the onset and end of the first phase:

- 1. Parents will rate their child's: (a) <u>Communication, Socialization and maladaptive behavior</u> using the Vineland Adaptive Behavior Scales (VABS-III; a structured interview); (b) <u>behavior</u> using the emotion dysregulation inventory (EDI) and the multidimensional assessment of disruptive behavior (MAP-DB); (c) <u>severity of core symptoms</u> using the autism impact measure (AIM); (d) <u>sleep habits</u> using the Children's Sleep Habits Questionnaire (CSHQ); (d) <u>health-related quality of life</u> of themselves using the Quality of Life in Autism Questionnaire (QOLA) Parent version; and (e) <u>gastrointestinal symptoms</u> the gastrointestinal symptoms a modified gastrointestinal sign and symptoms inventory (GISSI) and executive functions using the Behavior Rating Inventory of Executive Function (BRIEF).
- 2. Complete blood count (CBC), liver transaminases (LTs), and total bilirubin.
- 3. Plasma levels of 7-carboxy-CBD (the major circulating metabolite of CBD.
- 4. Possible biomarkers of treatment response (exploratory outcomes) including serum endocannabinoid (eCB) levels, relative mRNA expression levels of components of the eCB system in whole blood, RNA-sequencing of whole blood samples (transcriptome), plasma proteome, and gut microbiota

Additionally, at the end of the first phase physicians and caregivers will rate the global change in ASD-associated symptoms using the Overall Function Clinical Global Impression- Improvement (CGI-I) and the Caregiver Global Impression of Change (CGIC) assessments. Parents or primary caregivers will complete an Assessment of Blinding Questionnaire.

**Second phase:** Assessments at the end of the second phase will include: CGI-I and CGIC (global change in ASD-associated symptoms); adverse events; ABC-I, EDI, and MAP-DB (behavioral symptoms); SRS-2 and AIM (ASD core symptoms); CSHQ (sleep habits); BRIEF (executive functions), QOLA (quality of life); modified GISSI (gastrointestinal symptoms) and Assessment of Blinding Questionnaire.



Figure 3: Study design

### **Participants**

The study will be conducted at Shaare Zedek Medical Center, Jerusalem, Israel. Written informed consent will be obtained from a parent or legal guardian of participants after approval by the local institutional review board.

### <u>Inclusion criteria are</u>:

- Children aged 4 to 12 years.
- A diagnosis of ASD based on the Diagnostic and Statistical Manual of Mental Disorders [Fifth Edition; DSM-V], confirmed by CARS-2 assessment.
- Moderate or greater ASD-associated symptoms as measured by a rating of moderate or higher (≥4) on the Overall Function Clinical Global Impression—Severity (CGI-S).
- Aberrant Behavior Checklist-Irritability Subscale (ABC-I) score of 18 or higher.
- Social Responsiveness Scale 2<sup>nd</sup> edition (SRS-II) total score of 66T or higher.

### Exclusion criteria are:

- Bodyweight below 12.5kg or above or equal 57.5 kg.
- Current or past diagnosis of heart failure, drug addiction, schizophrenia, psychosis, bipolar disorder PTSD or MDD or diagnosis of schizophrenia in a first degree relative.
- A seizure or change in the antiepileptic medications in the 4 months prior to randomization.
- A physical exam and laboratory results are out of the normal range for individuals with ASD, including a significant impairment in heart, liver, or renal function.
- Any change in the pharmacological or behavioral treatment or change in the home or school settings (other than school holidays) in the 4 weeks prior to randomization or planned changes during the study.
- Cannabinoid treatment in the 4 weeks prior to randomization.
- Predicted low compliance to the study procedures (such as blood tests).
- Concurrent use of opiates or alcohol.

### Criteria for termination of participation:

- The Principal Investigator believes that continued participation endangers the participant.
- Upon a decision of the regulatory bodies: IRB or MOH.
- Upon request of one of the legal guardians

Terms for termination of participation: After termination of participation – participants will continue to receive the same treatments they received before termination, excluding the study treatment. These treatments will not be affected in any way by their decision to terminate their participation in the study

### **Procedures**

Screening: ASD diagnosis will be established using a structured assessment of DSM-5 criteria together with a Childhood Autism Rating Scale, Second Edition (CARS-2) total score ≥30. Caregivers will complete a medical history questionnaire covering demographic information, potential etiological factors (perinatal, genetic, imaging), comorbidities (epilepsy, allergies, immune-mediated disorders, sleep disturbances), autistic regression, diet, nutritional supplements, and behavioral treatments. Other assessments will include the CGI-S, ABC-I, SRS, and NVIQ (as detailed below). ADOS-2 - module, date and calibrated severity score will be documented. Blood samples- (15 ml) will be collected at 0 and 8 weeks.

- Complete blood count (CBC), liver transaminases (LTs) and total bilirubin will be measured as part of the safety analyses.
- Plasma levels of 7-carboxy-CBD<sup>62</sup> will be assessed to determine individual bioavailability of CBD. At 2-month, blood will be collected 3-4 hours post treatment administration.
- Serum endocannabinoids (ECs)<sup>16,19</sup> and relative mRNA expression levels (real-time PCR) of components of the eCB system in whole blood,<sup>16</sup> RNA-sequencing of whole blood samples (transcriptome),<sup>63</sup> and plasma proteome,<sup>64</sup> will be assessed to explore possible markers of treatment response.

### Stool samples will be collected at 0 and 8 weeks.

- Gut microbiota was demonstrated to be associated with ASD as well as symptom severity in multiple studies. 65-67

#### Study treatment:

Participants will receive terpenes-enriched CBD-predominant cannabis oil for oral administration (8.96 mg CBD and 0.32 mg THC per drop, T1/C28, <u>Bazelet</u>, Israel) or matched placebos: an oil with similar appearance, taste and smell for 8 weeks (first phase).

The target dose is: CBD-7.2mg/kg/d, THC-0.257mg/kg/d, and terpenes - 0.5mg/kg/d.

The initiation dose will be 0.1 drops/kg twice daily: morning and afternoon (6-9 hours apart) for 4 days (1.8mg CBD/kg/d); followed by 0.2 drops/kg twice daily (3.6mg CBD/kg/d) for 4 days and 0.4 drops/kg twice daily (7.2mg/kg/d) thereafter.

<u>Second phase:</u> At the end of the first 8-week phase participants will gradually stop the treatment they received in the first phase over 1 week: 0.2 drops/kg twice daily for 3 days; followed by 0.1 drops/kg twice daily for 4 days.

Participants who received placebo in the first phase will receive terpenes-enriched CBD isolate, and participants who received the study drug will continue with the same treatment for another 8 weeks.

The titration in the second phase will be like the first 8-week phase: at week 9: 0.1 drops/kg twice daily for 4 days (1.8mg CBD/kg/d); followed by 0.2 drops/kg twice daily (3.6mg CBD/kg/d) for 4 days and 0.4 drops/kg twice daily (7.2mg/kg/d) until week 17. At week 17, participants will gradually stop the treatment over 1 week: 0.2 drops/kg twice daily for 3 days; followed by 0.1 drops/kg twice daily for 4 days.

Based on previous studies the safety of the study treatment (in the target dose) is very high. If the LTs (at 0 or 8 weeks) will be between 2 to 3 times higher than the upper limits of the norm (ULN) we will not change the target doses and repeat the tests after 2 weeks. If the LTs are more than 3 times higher than the ULN we will decrease the target dose of the CBD by 50% and repeat the tests after 2 weeks. If the repeated LTs are less than 2 times higher than the ULN we will increase the daily CBD dose to 5mg/kg.

### Study visits

On-site visits: 4 visits: Screening (visit #1), Baseline (visit #2), 4 weeks (visit #3), 8 weeks (visit #4 - end of the first phase) and 17 weeks (visit #5 - end of the second phase). Phone visits to document compliance and adverse events: Three visits at study onset- (days 4, 8, and 12) and another 3 visits on weeks 6, 11, and 13. The PI may decide to hold the third meeting on Zoom

### **Outcomes and measures:**

### **Baseline evaluations (at screening):**

<u>Childhood Autism Rating Scale – Second Edition (CARS2)</u>. <sup>68</sup> CARS-2 is a validated tool for screening and classifying ASD, based on direct behavioral observation across 15 items (14 specific domains such as communication, body use, and response to stimuli, plus one global severity rating). Each item is scored from 1 (normal) to 4 (severely abnormal). Total scores of 30–36.5 indicate mild to moderate ASD, and scores >36.5 indicate severe ASD. The High-Functioning Form (CARS2-HF) is used for children ≥6 years with IQ >80, while the Standard Form (CARS2-ST) is used for all others.

Nonverbal Intelligence Quotient (NVIQ): NVIQ will be assessed using Raven's Colored Progressive Matrices (RPM), an untimed measure of problem-solving and abstract reasoning. The RPM consists of colored pattern sets (A, Ab, B) of increasing difficulty to assess observational and fluid intelligence. Test–retest reliability is typically >0.80. The RPM is generally considered to provide a more accurate estimate of NVIQ in children with ASD compared to the WISC or WPPSI.<sup>69-71</sup>

#### **Outcome Measures**

<u>ABC-I</u>: The ABC<sup>72,73</sup> is a caregiver-completed questionnaire with 58 items, organized into five subscales. The ABC-I (irritability) subscale consists of 15 items that measure the emotional and behavioral symptoms of ASD, including aggression toward others, deliberate self-injuriousness, temper tantrums, depressed mood and rapidly changing moods. The ABC-I has been accepted as the gold standard for measuring irritability in medication trials for ASD<sup>74</sup> and therefore, we will use it as the primary endpoint in this study. Individual items are rated from 0 (never a problem) to 3 (severe problem).

 $\underline{VABS-III}$  75: The VABS is a semi-structured caregiver interview designed to assess functional skills in three domains: Communication, Socialization, and Daily Living Skills. It also contains a short Maladaptive Behavior Domain. The Adaptive Composite Score estimates overall adaptive behavior. Vineland items are scored based on an open-ended question as 0 (behavior not performed), 1 (performed sometimes), or 2 (performed on a regular basis). The instrument provides Standard scores (mean = 100, SD = 15) and Age Equivalent scores

<u>SRS (Hebrew version)</u> <sup>76,77</sup>: The SRS is a 65-item caregiver or teacher questionnaire with five subscales: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Autistic Mannerisms. Items are rated on a 4-point Likert scale (0–3, total 0–195), with higher scores indicating greater impairment. Subscales yield T-scores; a Total T-score of 60–75 indicates mild to moderate impairment, and >75 indicates severe impairment. Caregivers will complete the SRS based on behavior during the previous 6 weeks. The SRS is widely used in ASD research. <sup>78-83</sup>

<u>CGI</u><sup>84</sup>: this is a 7-point scale designed to measure the severity of illness (CGI-S) and, an overall improvement from baseline (CGI-I). This measure has been used in many clinical trials in ASD.<sup>58,85,86</sup> Scores in the severity scale range from 1 (normal) through to 7 (amongst the most severely ill patients); in the improvement scale, scores range from 1 (very much improved) through 4 (unchanged) to 7 (very much worse).

<u>CGIC</u>: this is a 7-point scale designed to measure the overall improvement from baseline. This measure is completed by the primary caregivers and is similar to the CGI-I

<u>Autism Impact Measure (AIM)</u><sup>87,88</sup>: This is a 41-item caregiver-reported questionnaire designed to characterize core symptoms of ASD in individuals aged 3–18 years

<u>Multidimensional Assessment of Preschool Disruptive Behavior (MAP-DB)</u><sup>89</sup>: This 40-item caregiver-reported questionnaire assesses behavior across four domains: Temper Loss, Noncompliance, Aggression, and Low Concern for Others. It is available in three age-specific versions: 3-5 years, 6-8 years, and 9-10+ years.

<u>Emotion dysregulation inventory (EDI)</u><sup>90</sup>: This 30-item caregiver-reported questionnaire assesses observable signs of poor emotion regulation in children with autism.

<u>Behavior Rating Inventory of Executive Function (BRIEF)</u><sup>91</sup>: this is an 88 items Hebrew validated questionnaire, consists of 8 subscales, grouped into two index scores—Behavioral Regulation Index and Metacognition Index. Raw scores are converted into age- and sex-normed T scores.

<u>Children's Sleep Habits Questionnaire (CSHQ)<sup>92</sup></u>: this is a 33 items Hebrew validated questionnaire. A higher score reflects more significant sleep disturbances (range: 33–99, a score of  $\geq$ 41 classifies a "poor sleeper). The CSHQ has eight subscales: bedtime resistance; sleep onset delay; sleep duration; sleep anxiety; night waking; parasomnias; sleep-disordered breathing; and daytime sleepiness. This questionnaire has been used extensively in previous research in ASD

<u>Quality of Life in Autism Questionnaire (QOLA) – Parent version</u>. <sup>93</sup>The QOLA is a 48-item tool with two subscales to measure quality of life in parents of children with ASD. Part A (QoL subscale) includes 28 items assessing parents' overall quality of life, with scores ranging from 28 to 140 (higher scores indicate greater QoL). Part B (impact of ASD symptoms subscale) includes 20 items evaluating how problematic a child's ASD-related difficulties are for the parent, with scores ranging from 20 to 100 (higher scores indicate fewer problems).

<u>Modified gastrointestinal signs and symptoms inventory (GISSI)</u>: This 15-item questionnaire was adapted to this study based on the GISSI-17,<sup>94</sup> a brief parent-report screen for common gastrointestinal problems in children with ASD.

Adverse events (AE) will be monitored using a 31-item modification of the Dosage Record Treatment Emergent Symptom Scale. Recent health concerns, use of medical services, and change in study treatment dose and concomitant medications will be recorded as well. BMI, pulse rate, and blood pressure will be assessed at each clinic visit. Reports of new adverse events or worsening of previously reported events will be rated mild (present, but not persistent or requiring intervention), moderate (requiring intervention), or severe (posing a severe problem and requiring immediate intervention). Hospitalization will be documented as a serious adverse event. The PI will systematically evaluate all AEs for timing, biological plausibility, alternative causes, dose—response relationship, and prior knowledge to determine relatedness to the study drug, categorized as: not related, unlikely, possibly, probably, or definitely related.

### Table 1: Primary, secondary, and exploratory outcomes

**Primary outcome measure:** Change in the Aberrant Behavior Checklist-Irritability Subscale (ABC-I) score from Baseline to week 8.

#### **Main secondary outcome measures:**

- 1) Change from baseline to week 8 in the Vineland <sup>TM</sup> Adaptive Behavior Scales (VABS3)-Socialization Domain Score
- 2) Change from baseline to week 8 in the Social Responsiveness Scale (SRS-II) total raw score.

### Other secondary outcome measures:

- 1) Number of participants with severe, moderate, and mild treatment-emergent adverse events during the 8-week first phase.
- 2) Number of participants with clinically significant abnormal values in the CBC, liver transaminases, or total bilirubin or clinically significant abnormal values in the vital signs or physical examination at week 8
- 3) Change from baseline to week 8 in the BMI
- 4) Clinical Global Impressions-Improvement since baseline at week 8.
- 5) Caregiver Global Impression of Change (CGIC) since baseline at week 8.
- **6)** Change from baseline to week 8 in the Vineland <sup>TM</sup> Adaptive Behavior Scales (VABS3)-Communication and maladaptive behavior Domains Scores
- 7) Change from baseline to week 8 in the emotion dysregulation inventory (EDI)
- **8)** Change from baseline to week 8 in the multidimensional assessment of disruptive behavior (MAP-DB)
- 9) Change from baseline to week 8 in the autism impact measure (AIM).
- 10) Change from baseline to week 8 in the Quality of Life in Autism Questionnaire (QOLA) Parent version part A: parents' overall perception of their QOL- subscale score; and (c) part B: impact of ASD symptoms on parents' QOL- subscale score
- 11) Change from baseline to week 8 in the Children's Sleep Habits Questionnaire (CSHQ)
- 12) Change from baseline to week 8 in the gastrointestinal signs and symptoms inventory.
- 13) Change from baseline to week 8 in the Behavior Rating Inventory of Executive Function
- **14)** Global Impressions-Improvement since baseline at week 17
- 15) Caregiver Global Impression of Change (CGIC) since baseline at week 17.
- **16)** Change from baseline to week 17 in the Vineland <sup>TM</sup> Adaptive Behavior Scales (VABS3)-Communication and maladaptive behavior Domains Scores
- 17) Change from baseline to week 17 in the emotion dysregulation inventory (EDI)
- **18)** Change from baseline to week 17 in the multidimensional assessment of disruptive behavior (MAP-DB)
- 19) Change from baseline to week 17 in the autism impact measure (AIM).
- **20)** Change from baseline to week 17 in the Quality of Life in Autism Questionnaire (QOLA) Parent version part A: parents' overall perception of their QOL- subscale score; and (c) part B: impact of ASD symptoms on parents' QOL- subscale score
- 21) Change from baseline to week 17 in the CSHQ -total score
- 22) Change from baseline to week 17 in the gastrointestinal signs and symptoms inventory.
- 23) Change from baseline to week 17 in the BRIEF -Global Executive Composite (GEC) -T score

### **Exploratory outcomes**

- 1) Correlations between 'markers of CBD' at 8weeks (Plasma levels of 7-carboxy-CBD) and treatment outcomes, in the active treatment group.
- 2) Correlations between 'biomarkers' at baseline [markers of the endocannabinoid system, transcriptome, proteome, and gut microbiota] and treatment outcomes, in the treatment group.
- 3) Correlations between change in 'biomarkers' from baseline to 8 weeks and treatment outcomes, in the treatment group, in the placebo group, and in the entire cohort.
- 4) Correlations between 'child characteristics' at baseline [age, sex, level of function (DSM-5 levels of support required, CARS, VABS, CGI-S, ABC-I, SRS, NVIQ), etiological factors, comorbidities, history of autistic regression, diet, behavioral treatments and impact of high fever on social deficits status], and treatment outcomes, in the treatment group.
- 5) Correlations between 'child characteristics' at baseline and 'biomarkers' at baseline.
- 6) Effects of the treatment compared to placebo on 'biomarkers' change from baseline to week 8.
- 7) Correlations between plasma levels of 7-carboxy-CBD at 8 weeks and change in 'biomarkers' from baseline to 8 weeks, in the treatment group.
- **8)** Correlations between levels of 7-carboxy-CBD at 8 weeks, and 'biomarkers' at 8 weeks, in the treatment group.
- 9) Correlations between 'biomarkers' at baseline and levels of 7-carboxy-CBD at 8 weeks, in the treatment group.
- 10) Correlations among 'biomarkers' [markers of the endocannabinoid system, transcriptome, proteome, and gut microbiota]: at baseline (entire cohort), at 8 weeks (active treatment group, placebo group, and entire cohort), and when combining data from baseline and 8 weeks (entire cohort).
- 11) Correlations between each 'biomarker' and each behavioral assessment score (i.e., symptom severity) at baseline (entire cohort), at 8 weeks (active treatment group, placebo group, and entire cohort), and when combining data from baseline and 8 weeks (entire cohort).
- 12) Longitudinal changes in gut microbiota in the study group and in the placebo group and correlations with longitudinal changes in the behavioral assessments in these time points.
- 13) Cross-sectional correlations between gut microbiota and behavioral assessments at baseline (entire cohort) and at week 8 (active treatment group, placebo group, entire cohort) and when combining all time points (entire cohort).
- 14) Correlations between treatment outcomes in the placebo group ('placebo response') and the family characteristics: 'child characteristics' (age, IQ, severity of core symptoms, experience with previous oral treatments and perceived ability to understand the study goals) and 'parent characteristics' (age, education, and parental expectations and believes regarding pharmacological and natural treatments as assessed by the parental expectations and believes 29-item questionnaire).
- 15) Correlations between gut microbiota and gastrointestinal symptoms as assessed by the 30-item Health State Questionnaire (adverse events questionnaire) when combining all time points (entire cohort).
- 16) Correlations among all assessments including: 'treatment outcomes', 'child characteristics', and 'parent characteristics' (e.g., child QOL, parent QOL, severity of ASD symptoms, etc.).
- 17) Correlations between 'child characteristics', 'treatment outcomes', and 'biomarkers' assessed in this study, and polymorphism in genes that compose the endocannabinoid system and the 'methionine and methylation cycle' for participants in whom this data will be available (genetic assessments will not be performed as part of this study).

Table 2: Assessment Schedule during the first phase

| Visit Number | 1 | 2 | Cy. | € b | Cy. | 3 | Cy. | 4 |
|---|---|---|---|---|---|---|---|---|
| | Screening | Baseline | a | End of<br>Titration | c | 4W | d | 8W |
| Day Number (Visit Window) | -90 to 1 | 1 | 4±2 | 8±2 | 12±2 | 28±3 | 42±3 | 56±3 |
| Informed consent/assent | X | | | | | | | |
| Eligibility criteria <sup>§</sup> | X | X | | | | | | |
| Demographics & Medical history | X | | | | | | | |
| ASD criteria<br>- DSM-5 | X | | | | | | | |
| - CARS-2 | X | | | | | | | |
| Overall severity – CGI-S | X | | | | | | | |
| Behavioral problems: ABC-I | X | X | | | | X | | X |
| Core symptoms: SRS-2 | X | X | | | | X | | X |
| Nonverbal IQ | X | | | | | | | |
| Vital signs | X | X | | | | | | X |
| Physical exam (including BMI) | X | X | | | | | | X |
| Concomitant Medications | X | X | X | X | X | X | X | X |
| Parent expectations and believes | | X | | | | | | |
| Adverse Events | | X | X | X | X | X | X | X |
| Compliance with Intervention | | | X | X | X | X | X | X |
| Blood sampling* | | X | | | | | | X |
| Gut microbiota | | X | | | | | | X |
| Socialization – VABS-3 | | X | | | | | | X |
| QOLA; EDI; AIM | | X | | | | | | X |
| BRIEF, MAP-DB, GI problems | | X | | | | | | X |
| Sleep Habits – CSHQ | | X | | | | X | | X |
| Physician impression of overall change - CGI-I | | | | | | | | X |
| Caregiver impression of overall change – CGIC | | | | | | | | X |
| Assessment of Blinding<br>Questionnaire | | | | | | | | X |

<sup>§</sup> A diagnosis of ASD based on DSM criteria and CARS-2, core symptoms cannot be explained by the level of intellectual disability (NVIQ), age 4-12 years, weight 12.5-57.49 kg, CGI-S ≥4, ABCI-I score ≥18, SRS-2 total score ≥ 66, predicted compliance with study requirements including blood tests and tolerability to taste and smell of the study interventions.

<sup>\*</sup> CBC, liver transaminases, total bilirubin; Plasma levels of 7-carboxy-CBD; Serum endocannabinoid levels, relative mRNA expression levels of components of the eCB system in whole blood (real-time PCR), RNA-sequencing of whole blood samples, and plasma proteome.

Figure 4: Study Flow Chart

# **Study Outline**

Parents (and child when appropriate) are signed on the informed consent (and assent ) and than screened using the assessments defined in the inclusion criteria

Participant undergoes blood and stool sampling and physical examination A parent completes the ABC-I, SRS, AE, QOLA, CSHQ, mGISSI, EDI, BRIEF, MAP-DB, and AIM

A parent is interviewed to complete the VABS-3

Participant is randomised to either terpenes-enriched cannabinoids T1C28 or placebo compounds for 8 weeks

Participant undergoes the same evaluations as done in study onset A physician complete the CGI-I. A parent complete the CGIC Participant receive either terpenes-enriched cannabinoids T1C28 or terpenes-enriched CBD for a second 8-week period

Participant undergoes physical examination. A parent completes the ABC-I, SRS, AE, QOLA, CSHQ, mGISSI, EDI, BRIEF, MAP-DB, CGIC and AIM. A physician complete the CGI-I.

Data is monitored for accuracy Final data analysis- study completion

### **Statistical Analyses**

A detailed statistical plan is provided in the Statistical Analyses Plan (SAP).

Based on previously reported placebo effects on ABC-I scores in other ASD trials <sup>74,95,96</sup> and allowing for a slightly greater placebo effect due to higher expectations associated with cannabis treatment, we estimate that participants assigned to the placebo group will exhibit a mean 20% reduction from baseline ABC-I scores. Based on our preliminary results, we assume a small-to-medium effect size (0.35) for the study treatment—terpenes-enriched cannabis oil (T1/C28). Consequently, a sample size of 34 participants per group is required to achieve 80% power, using a mixed model of repeated measures (MMRM). To account for early withdrawals, an additional 15% will be recruited, resulting in a total of 39 participants per group.

This sample size is expected to provide sufficient power to detect differences in the primary outcome. However, an adaptive design with interim analysis by an external, non-blinded biostatistician will determine the final sample size.

For secondary and exploratory efficacy analyses, nominal p-values will be presented for informational purposes only.

The primary report will focus on odds ratios (OR) and 95% confidence intervals (CI). Additionally, a secondary analysis will evaluate the proportion of participants achieving the minimal clinically important difference (MCID) using a chi-square test or logistic regression analysis to compare proportions between groups. The analysis of the Vineland Adaptive Behavior Scales, Third Edition (VABS-III), will utilize Growth Scale Values (GSV), with adjustments for participants transitioning between age categories during the study.

All efficacy analyses will be based on an intent-to-treat (ITT) population, defined as all randomized subjects who receive at least one dose of the study medication and have post-baseline efficacy data available. For the primary efficacy outcome and key secondary outcomes, a perprotocol (PP) population will also be defined, consisting of ITT participants who substantially adhere to the study protocol.

The primary analysis assumes that ABC-I scores are missing at random (MAR), an assumption deemed reasonable for this study. Missing data are unlikely to differ systematically from observed values for unknown reasons.

The primary endpoint will be assessed using a Mixed Model for Repeated Measures (MMRM), implemented in SAS (PROC MIXED), R (lme4 package), or equivalent statistical software. Sensitivity analyses will include per-protocol analysis and may utilize multiple imputations to confirm the robustness of findings

Secondary analyses will be conducted using the same methodology as the primary ABC-I endpoint for each treatment sequence.

### **Data Management and Confidentiality**

<u>Identifiers</u>- We will use a mathematic manipulation on the participants' ID number (Xor with a 4-digit secret code) to assign a unique 'participant number'. We will use the participant number to avoid exposing personally identifiable information (PII). Only the Principal Investigator and data coordinating manager will have the list connecting the identified data with the participant number. The list will be kept in a locked desktop computer protected by two passwords and in a locked safe in Shaare Zedek Medical Center. Representatives of the IRB and MOH may have access to this identified list upon specific request.

<u>Confidentiality:</u> To protect the privacy of human subjects and maintain the confidentiality of study data we will use a strict separation between identified and non-identified data. <u>Identified data:</u> consent forms and contact information will not contain 'participant number'. It will be kept in a locked cabinet at Shaare Zedek Medical Center- SZMC. Electronic files of contact information and scans of consent forms will be kept in a locked desktop computer protected by two passwords.

ADOS-2 assessments (if performed) will be videotaped (with legal guardians' consent) to allow evaluation by two independent ratters. Files will be kept in external hard disks at a locked safe. All video files will be completely removed within 12 months after study completion. All other data, records, and biological samples will be captured and stored un-identified, using the participant number as the sole identifier.

Hard copies of all outcome questionnaires and assessment tools will be stored un-identified (participant number only) in locked cabinets at the study site (SZMC). Biological samples (sera, plasma, and stool samples) will be stored un-identified (participant number only) in locked freezers at the study site. Identified and non-identified data will be kept in different rooms. Only the study PI and the data coordinating manager will have access to study records, data, and specimens. Representatives of the IRB, and MOH are eligible to review study records.

<u>Data capture</u>, <u>verification</u>, <u>and disposition</u>: Study data will be captured using paper and pencil forms that will not contain identified data. Forms will be uploaded to the web application REDCap. REDCap is a secure web application for building and managing online surveys and databases. It can be used to collect any type of data including 21 CFR Part 11, FISMA, and HIPAA-compliant environments. REDCap supports online and offline data capture for research studies and the REDCap Consortium is composed of thousands of active institutional partners in over one hundred countries.

All data (hard copy and electronic) will be stored for 15 years.

<u>Sharing study results:</u> The results of all baseline assessments (CARS-2, nonverbal IQ), blood work, and other data regarding study participation (including study assignments and individual results) will be shared with the primary care providers.

### **Procedures Description:**

The principal investigator (PI) for the clinical investigation is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported in the eCRFs and in all other reports during the clinical investigation

The Site Clinical Coordinator for the clinical investigation is responsible for:

1 Maintaining all of the study-related files: This includes maintaining all logs such as:

- Ethics Approvals and all communications with the ethic committees (such as protocol amendments and serious adverse events reports)
- Protocol Deviation Log
- Subject Informed Consent (SIC) Signature Log
- Investigation Team Log
- 2 Correct filling of the eCRFs based on source documentation and live documentation
- 3 Maintaining contact with study subjects, and coordinating study visits

At the start of the clinical study, the Clinical Coordinator will make sure that all study files for the following:

- IRB/EC/Helsinki Committee Documents.All IRB Correspondence is on file. The study staff are IRB approved prior to performing any study procedures. Adverse events and deviation procedures for reporting to IRB per current guidelines are in place. All versions of the IRB protocols and informed consent forms are on file. Signed Good Clinical Practice compliance form, financial disclosure and CV for the PI and sub investigators.

#### Other documents:

- CVs for all study staff are on file and updated within the last 2 years
- Medical licenses for the Sub-Investigators are on file and updated prior to the expiration
- Delegation Log is updated and procedures for updating the log with new staff are in place
- All other essential documents have been prepared and completed as appropriate

Before, during, and at the close of the study period, study documentation will be monitored by the Clinical Coordinator for the following:

- Informed Consent Form (ICF)
  - o Ensure that subject identification is on all pages of the ICF, if applicable
  - o Documentation of subject receiving a copy of the consent form is present
  - o Clinic note documents informed consent process
  - The parents or a legal guardian of the subject and study representative signed and dated the consent form for their self
  - O Note to file completed for any informed consent deviations.
  - o Ensure a valid (current version date) copy of the consent form was used

#### **Protocol**:

- Confirm that the study staff is conducting the study in compliance with the protocol approved by IRB/CE/Helsinki Committee and are trained in Good Clinical Practices (GCP).
- The protocol deviations (exceptions and violations) are documented in the subject chart and reported to IRB/CE/Helsinki Committee as required.
- Ensure any deviations are logged in the form 'Protocol Deviations'

### **Source Documents:**

- Review subject charts to ensure accuracy, completeness, and legibility of the data
- Any correction made to the source documents is dated, initialed, and explained. The original entry should not be obscured.
- The protocol-specific source documents are on file.
- Source documents are completed in ink or electronically.
- Note to files are generated for missing or incomplete data, and to explain any discrepancies or additional comments.

### **Case Report Forms:**

- Ensure that the data reported on the CRF is consistent with the source documents.
- Discrepancies between the source documents and eCRF are explained in a note to file or captured in a comment in the eCRF.

### **Biological samples**

Biological samples will be labeled with participant numbers and stored in locked freezers. The legal guardians will decide in the consent form if the samples will be kept after the termination of the study for possible use in further studies or be destroyed upon termination of the study.

### **Blood samples**

Blood (6 ml in tubes with procoagulant, 6 ml in tubes with EDTA, and 3 ml in Tempus<sup>™</sup> Blood RNA Tube) will be collected at the baseline (9-11 AM) and at 2-month (on 9:00- 11:00 AM, 3-4 hours post treatment administration).

Assessments will include:

- Plasma levels of 7-carboxy-CBD
- Serum endocannabinoid levels
- Relative mRNA expression levels of components of the eCB system (CB1R, CB2R, NAPE-PLD, FAAH, DAGL, and MAGL) normalized to GAPDH in whole blood.
- RNA-sequencing of whole blood samples (transcriptome), and plasma proteomics will be performed pre and post-treatment to discover treatment-responsive biomarkers which correlate with behavioral improvement.

### Stool samples

Stool samples will be collected using OMNIgene GUT sample collection kit (DNA Genotek, Canada). This kit homogenizes the sample and stabilizes the DNA for up to 60 days at room temperature. Participants will receive the kits in advance: a first kit during the screening visit, a second kit during the 2<sup>nd</sup> or 3<sup>rd</sup>. Participants will be instructed to use the kits within 2 weeks prior to their next visit (baseline, 8 weeks) and bring them with them to the next visit. Stool samples will not be collected if the participant had received any antibiotic treatment during the 4 weeks prior to the sampling day. Any antibiotic treatment, special diets, and use of probiotics during the 4 to 8 weeks prior to the sampling day - will be documented.

### **Informed Consent Process**

Subjects' legal guardians interested in having their children participate in the clinical investigation will be screened by the participating physician.

Subjects' legal guardians will then be given a copy of the Patient Informed Consent with ample time to read and review the document and ask questions before signing.

Subjects will meet with one of the investigators to discuss investigational participation and any questions they may have regarding the investigation, the investigational device, and the informed consent.

The informed consent will be signed by the legal guardian, during the meeting with one of the participating investigators.

A photocopy of the signed patient informed consent form will be provided to the legal guardian prior to the procedure.

Subjects requesting to withdraw consent will be disqualified from the investigation at no cost or consequence

All subjects in this study are pediatric subjects (4-12) with ASD and are therefore unable to sign an informed consent. A legal guardian will sign the informed consent. Assent form will be obtained from any participant who is able to give it.

### **Vulnerable Population**

This clinical investigation will be conducted on pediatric (4-12 years old) ASD populations. Vulnerable patients' legal guardians will be responsible for patient informed consent.

### Data and Safety Monitoring Board (DSMB)

An independent Data and Safety Monitoring Board (DSMB) will oversee the conduct of the trial. The DSMB is responsible for monitoring study progress, including data quality, recruitment, retention, and the overall risk—benefit balance. It will also consider external developments relevant to participant safety and research ethics. The DSMB will review interim analyses as needed, although no formal stopping rules are defined for this study, and will ensure that all trial data remain confidential. The DSMB will provide regular reports to the Bazelet Group regarding participant safety and trial progress, and will make recommendations on whether the study should continue as planned, be modified, or be terminated. In addition, the DSMB will advise the Bazelet Group on issues related to study conduct, enrollment, or data integrity. The DSMB will conclude its responsibilities upon completion of follow-up for the final participant.

### Randomization and blinding

Eligible subjects will be assigned an enrollment number in sequential order beginning with 01. Allocation to the treatment arm will be based on a randomization list. A randomization scheme will be generated by an external unblinded biostatistician. The blocked randomization will be performed using SAS statistical software V9.4 via the plan procedure with a fixed block size. The randomization scheme and lists will be sent to the study site. The randomization list will include sequential numbers and assigned 4-letter codes. Randomization will be kept at a 1:1 ratio. The randomization list will be encrypted by password and will be sent prior to first dosing to the principal investigator.

The study active treatments as well as the placebo treatments will be packed in similar bottles and packages and will have similar appearance, taste, and smell.

CBD-predominant cannabis oils and matched placebo will be prepared, bottled, and labeled by the Bazelet Group (Or Akiva, Israel). CBD, terpenes, and THC (when applicable), together with a taste and odor mixture, will be dissolved in olive oil to yield a concentration of 28% CBD (280 mg/g, equivalent to 256 mg/mL, or 8.96 mg per 0.035-mL drop) and 9 mg THC/mL (0.32 mg per 0.035-mL drop). An international company (dsm-firmenich) designed the taste and odor mixture to ensure that all three treatments (study drug, terpene-enriched CBD oil, and placebo) are indistinguishable.

The code key for the active/ placebo labels will be kept by the external biostatistical until study-end. Neither the principal investigator nor any other team member or individual will have access to the codes until study-end.

To assess the blinding state, caregivers, participants (when applicable) and researchers will complete an Assessment of Blinding Questionnaire at the end of the randomized study.

### **Study Interventions**

CBD-predominant cannabis oil (CBD 3.6 mg/kg twice daily; THC 0.128mg/kg twice daily, and terpenes 0.25mg/kg twice daily) will be administered orally **as an add-on** to any existing treatment.

#### **Dose Justification**

The target dose of 7.2mg CBD/kg/d and 0.257mg THC/kg/d divided into 2 daily doses is based on the results of the randomized study that was completed recently<sup>50</sup> in which the target dose was 10mg CBD/kg/d and 0.5mg THC/kg/d and on our clinical experience in recent years in more than 400 children. Notably, ongoing clinical trials of CBD for children with ASD use 3-20mg/kg/d, and most are using 10mg/kg/d.<sup>51</sup> The safety of plant-derived CBD isolate at doses of 10-50mg/kg/d was demonstrated in multiple placebo-controlled studies in children with epilepsy and lower doses are associated with fewer AEs.<sup>97-101</sup> At a dose of 7.2mg/kg/d we expect no treatment related adverse events.

### Administration

CBD rich oil will be administered by drops containing 0.035 ml / 8.96 mg CBD each. The CBD dose will be up-titrated over 8 days:

Days 1-4: 0.1 drops per Kilogram of Bodyweight (rounded number)— twice daily (1.8 mg/kg/d) Days 5-8: 0.2 drops per Kilogram of Bodyweight (rounded number – twice daily (3.6 mg/kg/d) Days 9-56: 0.4 drops per Kilogram of Bodyweight (rounded number – twice daily (7.2 mg/kg/d)

The CBD dose will be down-titrated at the end of the randomized study over 7 days: Days 57-60: 0.2 drops per Kilogram of Bodyweight (rounded number – twice daily (3.6 mg/kg/d) Days 61-64: 0.1 drops per Kilogram of Bodyweight – twice daily (1.8 mg/kg/d)

On day 65, the parents or legal guardian will decide if the treatment will be discontinued or be switched to a second treatment (either terpenes enrich CBD isolate or CBD-predominant oil) at the same dose for 4 days followed by 0.2 drops per Kg X 2/d for another 4 days and 0.4 drops/kg X2/d until the end of the second phase.

### **Amendments to the Protocol**

The study coordinator will ensure that

- 1 Amendments to the Clinical Investigation Plan are documented, using the form 'Amendment and Revision Sheet'
- 2 Approval is documented, using form 'Clinical Investigation Document Approval Log'' The amended protocol is sent to all investigators and the EC/IRB/Helsinki Committee after approval

### **Deviations from the Protocol**

Neither the Principal Investigator nor any of the sub-investigators are authorized to deviate from the protocol, except as specified in 4.5.4 b of ISO 14155:2011 and 21 CFR 812.150 (a)(4), specifically requests for deviations, and reports of deviations, if the deviation affects subject's rights, safety, and wellbeing, or the scientific integrity of the clinical investigation. Under emergency circumstances, deviations from the protocol to protect the rights, safety, and well-being of human subjects may proceed without prior approval of the sponsor and the EC/IRB/Helsinki Committee. Such deviations shall be documented and reported to the sponsor and the EC/IRB/Helsinki Committee as soon as possible.

The research coordinator will prepare the EC/IRB /Helsinki Committee Notifications letter using the EC Notification Form if any reportable serious deviations or adverse events were recorded and send them to the Ethics Committee/Institutional Review Board/Helsinki Committee and Principal Investigator, according to this protocol.

All notifications will be carried out within the time frames specified by local regulatory authorities.

### **Statements Of Compliance**

- 1 This clinical investigation will be conducted in accordance with ethical principles stated in the Declaration of Helsinki and in compliance with all national and local regulatory requirements for the safety and protection of human subjects.
- 2 This clinical investigation will be implemented only upon receiving all final notification/authorizations from local and national regulatory and Helskinki/EC/IRB authorities, as appropriate.
- 3 This clinical investigation will comply with any additional requirements set forth by the Helsinki/EC/IRB and/or regulatory authorities.
- 4 This clinical investigation provides clinical study medical insurance for study participants as required by local and national regulatory authorities.
- 5 This protocol was written in accordance with the ISO 14155:2011 Standard for Clinical investigation of medical devices for human subjects Good Clinical Practice

### **Early Termination or Suspension of the Clinical Investigation**

Grounds for suspension or premature termination of the clinical investigation include but are not limited to:

- Non-compliance of the investigational site personnel to the protocol and or investigational procedures
- Serious Adverse Events that demonstrate danger to the patient population
- Unethical performance on the part of any of the investigators
- Failed audit of investigation with serious flaws to study design, performance or outcomes
- Business/Financial issues that cannot be resolved
- Other unforeseen events that give the PI reasonable doubts to the safety of the participants which cannot be resolved in a reasonable time

#### **Publication Policy**

The results of this clinical investigation may be published in a mainstream peer-reviewed professional journal as per Chapter I. of the agreement between the Shaare Zedek Medical Center and the Sponsor

#### **Adverse Events**

An **adverse event** is any undesirable or unintentional or unexpected event (sign, symptom, illness, abnormal laboratory value, or other medical events) that occurs during the course of the study, whether or not considered related to the study interventions. This definition includes events related to the investigational treatments and also includes events related to the procedures involved.

Regardless of the relationship to the investigational treatments, all moderate to serious adverse events occurring from the time that the informed consent is signed must be recorded in the patient's CRF.

A **mild adverse event** is one that the symptom does not influence performance, require drug treatment or prevent the patient from carrying on with normal life activities.

A **moderate adverse event** is one that the symptoms make the patient uncomfortable and causes some impairment to normal life activities and require treatment for symptom(s).

A **serious adverse event** is an adverse event that:

- Led to death
- Led to a serious deterioration in the health of the subject, that either resulted in
  - o A life-threatening illness or injury, or
  - o A permanent impairment of a body structure or body function, or
  - o In-patient or prolonged hospitalization, or
  - Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function

In the event of an emergency resulting from the clinical investigation, all emergency treatment will be provided at no cost to the patient. Clinical Investigation Insurance has been provided to ensure all costs be covered if necessary.

The principal investigator will notify the sponsor immediately (within 24 hours) of any serious adverse event. All reports to the appropriate authorities will be made by the principal investigator as set forth in the standard clinical practices outlined in the 21 CFR (§ 812.150(a)(1), § 812.46(b) and § 812.150(b)(1))/ MEDDEV 2.7/3 Dec 2010 and ICH-GCP Guidelines.

Adverse Events will be reported and treated as per the standard clinical practices outlined in the 21 CFR (§ 812.150(a)(1), § 812.46(b) and § 812.150(b)(1))/ MEDDEV 2.7/3 Dec 2010 and ICH-GCP Guidelines

Anticipated adverse events include rare insomnia, irritability, and intolerance of the taste and smell.

# Appendix 1 – non-generic questionnaires

The Hebrew version of the following questionnaires appears in the investigator brochure.

| Demographics and medical history questionnaire | 31 |
|------------------------------------------------|----|
| Health State Questionnaire (adverse events) | 34 |
| Parental expectations and beliefs | 35 |
| Assessment of Blinding Questionnaire | 36 |
| Gastrointestinal signs and symptoms inventory | 37 |

# Cannabinoid treatment in children with ASD – Demographic questionnaire

| e: _ | GUID: | Informant: Mothe / Father / Guardian |
|---|---|---|
| 1. | Please describe at which age and | /her development or communication? No/Yes the nature of the regression: |
| 2. | When your child has a high ten | nperature, does she/ he have a substantial n? No/Yes (Please specify) |
| 3. | Has your child had a genetic te<br>CMA (chip) - No/Yes /unknown | sting? No/Yes<br>a; Exome sequencing - No/Yes /unknown |
| 4. | Does your child have a genetic | diagnosis? No/Yes |
| 5. | Angelman syndrome, or substant | yndromic ASD? (Such as Down syndrome or tial deficits in motor function or cardiac problems, or s (Please specify |
| 6. | | or an uncle with ASD (even mild)? No/Yes (Please |
| 7. | | or an uncle with intellectual disability? No/Yes |
| 8. | Birth week:: Normal | / 35-36/ 32-34/ 29-31/23-28 |
| 9. | Birth weight: Small for Gestational age/ Larg | Appropriate for Gestational Age / ge for Gestational age |
| 10. | Curse of delivery: Normal / Ces | arean / Vacuum/ Forceps, APGAR: |
| 11. | • | NICU after the labor? No / Yes-less than 24 hours / onger than 4 weeks |
| 12. | Was you child ever hospitalize | d in ICU: No/Yes (Please specify) |
| 13. | accident in the first two years of | a pregnancy or childbirth or a serious illness / of life? (Severe complications of prematurity, mening ospitalization in intensive care, drowning or suffocation |
| 14. | How old was your child when h | ne was first diagnosed with ASD? |
| | | ne/she started attending a special education progra |

| 16. | Did your child suffer (for more than 6 months) from any of the following problem (Please mark all that applies) | s? |
|---|---|---|
| | Significant behavioral difficulties / Anxiety/ Significant sleep disorder / ADHD / Epilepsy / High sensitivity to noise, smell or touch /Unusual seeking of stimulations: smell, touch, sight / Low motor skills / GI problems / Food allergy / Food sensitivity | |
| 17. | Does your child have any other chronic diseases? No/Yes | |
| 18. | Has your child ever taken any medications on a regular basis (for more than a month)? No/Yes (Please mark all that applies) | |
| | Antipsychotics: Neuleptil (Pericyazine) / Rispond, Risperdal (Risperidone) / Abilify, Ariply (Aripiprazole) / Entumine (Clothiapine) / Zyprexa (Olanzapine) / Promethazine (Prothiazin) / Seroquel (quetiapine) / Ziprasidone (Geodon) / Nozinan (levomepromazine) / clozapine | • |
| | Stimulants: Ritalin, Concerta, Focalin / Attent, Vyvanse | |
| | SNRI: Atomic, Strattera | |
| | alpha-2 agonists: Clonirit (clonidine), Intuniv (Guanfacine) | |
| | Mood stabilizers: Depalept (Valproic acid) / Tegratol, Timonil (Carbamazepine) | |
| | Benzodiazepines: Rivotril, Clonex (Clonazepam) / Xanax (alprazolam) | |
| | <b>SSRIs</b> : Cipralex, Lexapro (escitalopram), Prozac, Prizma, Flutine (fluoxetine), Favoxil (fluvoxamine), Seroxat (paroxetine), Lustral, Serenada, Zoloft (sertraline) | |
| | Other: | |
| 19 | Is your child currently taking any medications on a regular basis? No/Yes | |
| 1.N<br>2 N | Name: daily dose since<br>Name: daily dose since | |
| 3.N | Name: daily dose since | |
| 4.N | Name: daily dose since | |
| 5.N | Name: daily dose since | |
| 20. | Has your child ever taken any nutritional supplements (for more than a month)? No/Yes (Please mark all that applies) | |
| | Vitamins: Folic Acid / Folinic Acid / B12 / B6 / Vitamin D<br>Minerals: Magnesium / Iron / Calcium | |
| | Other: Carnitine (L-carnitine, Acetyl carnitine) / Sulforaphane, Glucoraphanin Other: Melatonin / Probiotics/ Omega – 3 Other: | |
| 21. | If any of the mentioned nutritional supplements were discontinued in the past 3 months, please specify which and when: | |
| 22. | Has your child received antibiotics in the past two months? No/Yes (Please specify Name, daily dosage and for how long) | |

| 23. | Ha | s your chi | ld currently taking | any nutrition | al suppleme | ents? No/Yes | |
|---|---|---|---|---|---|---|---|
| 1.N | am | e: | dail | y dose | since | · | |
| | | | dail | | | | |
| 3.N | am | ie: | dail | y dose | dose since | ee | |
| 4.N | am | ıe: | dail | y dose | since | | |
| 5.N | am | ie: | dail | y dose | since | 2 | |
| | chi | ild consum | y the amount of cow<br>es per day:<br>o to half a glass / abou | ` | | , | · |
| | Lo | w Carbs (n | currently on a speci<br>nodified Atkins) | · | | | |
| | No | Y es (Pleas | se specify Which and | for now long | ) | | |
| 26. | На | as your chi | ild ever taken medic | cal Cannabis | / CBD / Car | nabis products? | |
| | No | /Yes (Pleas | se specify for how los | ng he/she took | t it and wher | was it discontinued | l) |
| | 1. | | Medical Cannabis wl<br>months. Discontin | • | | · | 8:1) |
| | 2. | for | Cannabis which most months. Disconti | nued | years and | dmonths ago. | ŕ |
| | 3. | Other: | months. Disconti | | | | |
| | | for | months. Disconti | nued | years and | d months ago. | |
| | | - | currently receiving | | | | |
| | 1. | | | Hours per | r week: | Since | |
| | 2. | | | Hours per | . week: | Since | |
| | <i>3</i> . 4. | | | Hours per | r week: | Since | |
| | 4.<br>5. | | | Hours per Hours per | rweek: | Since | |
| | | ease specify | y all the schools/ edu | | | | |
| | Ag | ge | Program: | | | | |
| | Ag | ge | Program: | | | | |
| | Ag | ge | Program: | | | | |
| | | | Program: | | | | |
| | Ag | ge | Program: | | | | |
| | Ag | ge | Program: | | | | |
| | Ag | ge | Program: | | | | |
| 29. | Pai | rents educ | ation (years): Moth | er: | | Father: | |
| 30. | Pai | rents occu | pation: Mother: | | Fat | ther: | |

| 1 | | _ | Sometimes | Always | mild | moderate | Severe | Treatment related |
|---|---|---|---|---|---|---|---|---|
| | Dizziness | | | | | | | |
| | Drowsiness | | | | | | | |
| | Restlessness | | | | | | | |
| | Aggression | | | | | | | |
| | Increased tantrums | | | | | | | |
| | Emotional liability | | | | | | | |
| | Hair loss | | | | | | | |
| | Rash | | | | | | | |
| | Blurred vision | | | | | | | |
| | Nausea | | | | | | | |
| | Vomiting Abdominal pain | | | | - | | | |
| | Concentration problem | | | | | | | |
| | Dry mouth | | | | | | | |
| | Tremors | | | | | | | |
| | Headache | | | | | | | |
| | Insomnia | | | | | | | |
| | Involuntary movements | | | | | | | |
| | Depression Depression | | | | | | | |
| | Memory problems | | | | | | | |
| | Constipation | | | | | | | |
| | Loss of appetite | | | | | | | |
| | Gain of appetite | | | | | | | |
| | Diarrhea | | | | | | | |
| | Nasal congestion | | | | | | | |
| | Sweating | | | | | | | |
| | Weakness | | | | | | | |
| | Increased salivation | | | | | | | |
| | Increased anxiety | | | | | | | |
| | Confusion | | | | | | | |
| 31 | Suicidal thoughts | | | | | | | |

# Parental expectations and beliefs

The following table presents various statements. Please indicate to what extent do you agree with each statement (your answers will have no effect on your participation in the study)

| # | Statements | Strongly<br>Agree | Quite agree | Not so agree | Not at all agree |
|---|---|---|---|---|---|
| 1 | When I give my child medicine (for example to relieve pain) he/she usually understands | | | | |
| _ | that the treatment may help him/her. | | | | |
| 2 | My child can understand that the treatment given in the study may improve his / her | | | | |
| | behavior. | | | | |
| 3 | My child can understand that the treatment given in the study may improve his / her communication difficulties. | | | | |
| 4 | My child's condition in the last month is worse compared to his average condition | | | | |
| 5 | It is hard for me to deal with my child's behavioral difficulties (I am losing patience) | | | | |
| 6 | When I am calm and patient my child is usually calmer too | | | | |
| 7 | I believe that the treatment given in the study may <b>greatly</b> improve my child's communication difficulties. | | | | |
| 8 | I believe that the treatment given in the study may <b>greatly</b> improve my child's behavioral difficulties | | | | |
| 9 | I personally know a family that treatment similar to the one given in the study - helped her a lot. | | | | |
| 10 | In the last year, my child received natural or medicinal therapy that helped him/ her with his/ her behavioral difficulties. | | | | |
| 11 | In the last year, my child received natural or medicinal therapy that helped him/ her with his/ her communication difficulties. | | | | |
| 12 | In the last year my child received natural or medicinal treatment for the behavioral difficulties which was discontinued due to side effects | | | | |
| 13 | My child is relatively sensitive to side effects of medications | | | | |

# Questions for the child participating in the study

| ☐ What do you see in the picture? |
|---|
| ☐ Why do you think the child is taking medicine? (Maybe his tummy hurts and they want to help him feel better, maybe he |
| has trouble behaving nicely and they want to help him) |
| ☐ How can the medicine help the child? |
| ☐ Do you sometimes have trouble behaving nicely? |
| ☐ We want to give you a treatment that will help you feel calmer and behave more nicely. Do you think that will help you? |
| ☐ We also believe the treatment can help you with your communication, like talking, understanding, and playing with others |
| Do you think that will help you? |
| Rank (from 1-10): |
| A. The child's ability to understand that the medicine given to him will improve his behavioral difficulties |
| B. The child's expectations that the treatment will help with his behavior problems |

# **Assessment of Blinding Questionnaire**

- 1) Please select the option that best reflects your beliefs regarding the treatment that your child received in the study:
  - A) I am convinced that the treatment was 'real treatment'
  - B) It seems to me that the treatment was 'real treatment'
  - C) It seems to me that the treatment was 'placebo'
  - D) I am convinced that the treatment was 'placebo'
  - E) I really do not know

| 2) | If you chose A, B, C, or D, please tell us why you chose this option (you can choose more than one option) |
|---|---|
| | A) Due to the appearance, smell, or texture of the treatment. please specify: |
| | B) Due to the effectiveness of the treatment |
| | C) Due to the inefficiency of the treatment |
| | D) Due to the side effects of the treatment. Please indicate which side effects: |

E) I have such a feeling but I cannot point to the reason

# Gastrointestinal signs and symptoms inventory (modified GISSI-17)

| Partic | cipant research ID | | | |
|---|---|---|---|---|
| Your r | relationship to this child: Mother Father Other: | | | |
| | of the questions on this form are about THE LAST S put a check (V) in the box that best describes your c | | S. | |
| | last 6 weeks, has your child experienced any of the foll | owing gast | rointestina | l (tummy) |
| sympto | oms: | Yes | No | Unsure |
| 1.<br>2. | Abdominal (belly) pain<br>Nausea | | | |
| 3. | In the last 6 weeks, how often did your child usually a Less than once a week b 1-2 times a week c 3-6 times a week d Once a day e 2-3 Times a day f More than 3 times a day g Unsure | have BMs? | | |
| 4. | In the last 6 weeks, what were your child's BMs usual a. Very hard b. Hard c. Not too hard and not too soft d. Very soft or mushy e. Watery f. Unsure | illy like? | | |
| | In the last 6 weeks, did your child: | Yes | No | Unsure |
| 5.<br>6. | Appear to feel pain when having a BM? Have to rush to the bathroom for a BM? | | | |
| | In the last 6 weeks, has your child: | Yes | No | Unsure |
| 7. | Spit up $\geq 2x$ per day? | | | |
| 8. | Experienced retching? | | | |
| 9. | Tilted his/her head to the side and arched back? | | | |

| Clinical Protocol 0336-24-SZMC |
|-----------------------------------|
| Terpenes-enriched cannabis in ASD |

September 1, 2025, Version 3.0 Confidential and Proprietary

| In the last 6 weeks, has your child missed activities due to: | Yes | No | Unsure |
|---|---|---|---|
| 10. pain and/or discomfort? | | | |
| 11. Vomiting | | | |
| 12. problems with BMs | | | |
| 13. <u>In the last 6 weeks</u> , did your child push his abdomen with his his/her abdomen against or lean forward over furniture? | s/her hands | or your ha | nds, push |
| 14. <u>In the last 6 weeks</u> , did your child choke, gag, cough, or sour swallowing or with meals? | nd wet durin | ng or after | |
| 15. <u>In the last 6 weeks</u> , has your child started to refuse many foo the past? | ds that he o | r she wou | ld eat in |

Appendix 2

Placebo-controlled clinical trials of cannabinoid therapy in ASD with published results

| Study | Treatment | Target daily | Participants | Primary Key Secondary | | Results |
|---|---|---|---|---|---|---|
| | | dose | & design | outcome/s | outcomes | |
| Aran et | CBD-rich cannabis | 10mg CBD | N=150; age | Behavioral | 1. Social | Both cannabinoids |
| al. [ <sup>50</sup> ] | extract, 1 CBD:THC | per kg of | 5-21 years; | improvement at | Responsiveness | were superior to |
| | ratio = 20:1; | body weight, | Cross-over; | week 12: | Scale (SRS-2) | placebo in 2 out of 4 |
| | Pure CBD&THC, <sup>2</sup> | divided into 3 | Two 12- | 1. CGI-I <sup>3</sup> | 2. Autism Parental | assessments: CGI-I <sup>3</sup> |
| | CBD:THC = 20:1 | daily doses | week periods | 2. HSQ-ASD <sup>4</sup> | Stress Index (APSI) | and SRS-2. No severe |
| | | - | _ | | 3. Safety | adverse events |
| Silva et | CBD-rich cannabis | Variable dose: | N=60; age 5- | Primary Vs Secondar | Primary Vs Secondary outcomes were not | |
| al. [102] | extract 5 CBD:THC | 1.0-11.6 mg | 11 years; | specified. <b>1.</b> A semi-structured interview | | in 3 out of 9 |
| | ratio = 9:1 | CBD ( <u>total</u> ) | Parallel | prepared by the authors. 2. Autism | | symptoms assed by |
| | | divided into 2 | groups; | Treatment Evaluation Checklist (ATEC). | | the interview but not |
| | | daily doses | 12 weeks | <b>3.</b> Childhood Autism Rating Scale (CARS) | | on ATEC or CARS |

<sup>&</sup>lt;sup>1</sup> BOL-DP-O-01-W, a whole-plant cannabis extract containing CBD and THC at a 20:1 ratio

<sup>&</sup>lt;sup>2</sup> BOL-DP-O-01, purified CBD + purified CBD at a 20:1 ratio

<sup>&</sup>lt;sup>3</sup> CGI-I: Clinical Global Impression-Improvement was used to measure improvement in disruptive behaviors by incorporating anchoring instructions related to behavioral difficulties.

<sup>&</sup>lt;sup>4</sup> HSQ-ASD: Home Situations Questionnaire-ASD, a parent-rated measure of noncompliant behavior in children with ASD

<sup>&</sup>lt;sup>5</sup> CBD-rich cannabis extract containing CBD and THC at a 9:1 ratio, supplied at a very low concentration (5mg/mL) by the Associação Brasileira de Apoio Cannabis Esperança (ABRACE)

# References

- 1. Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. *Lancet*. Aug 11 2018;392(10146):508-520. doi:10.1016/s0140-6736(18)31129-2
- 2. Goel R, Hong JS, Findling RL, Ji NY. An update on pharmacotherapy of autism spectrum disorder in children and adolescents. *Int Rev Psychiatry*. Feb 2018;30(1):78-95. doi:10.1080/09540261.2018.1458706
- 3. Scahill L, Jeon S, Boorin SJ, et al. Weight Gain and Metabolic Consequences of Risperidone in Young Children With Autism Spectrum Disorder. *J Am Acad Child Adolesc Psychiatry*. May 2016;55(5):415-23. doi:10.1016/j.jaac.2016.02.016
- 4. Tesfaye R, Wright N, Zaidman-Zait A, et al. Investigating longitudinal associations between parent reported sleep in early childhood and teacher reported executive functioning in school-aged children with autism. *Sleep*. Sep 13 2021;44(9)doi:10.1093/sleep/zsab122
- 5. Reynolds AM, Soke GN, Sabourin KR, et al. Sleep Problems in 2- to 5-Year-Olds With Autism Spectrum Disorder and Other Developmental Delays. *Pediatrics*. Mar 2019;143(3)doi:10.1542/peds.2018-0492
- 6. Suraev AS, Marshall NS, Vandrey R, et al. Cannabinoid therapies in the management of sleep disorders: A systematic review of preclinical and clinical studies. *Sleep Med Rev*. Oct 2020;53:101339. doi:10.1016/j.smrv.2020.101339
- 7. Kaul M, Zee PC, Sahni AS. Effects of Cannabinoids on Sleep and their Therapeutic Potential for Sleep Disorders. *Neurotherapeutics*. Jan 2021;18(1):217-227. doi:10.1007/s13311-021-01013-w
- 8. Spanagel R, Bilbao A. Approved cannabinoids for medical purposes Comparative systematic review and meta-analysis for sleep and appetite. *Neuropharmacology*. Sep 15 2021;196:108680. doi:10.1016/j.neuropharm.2021.108680
- 9. Schnapp A, Harel M, Cayam-Rand D, Cassuto H, Polyansky L, Aran A. A Placebo-Controlled Trial of Cannabinoid Treatment for Disruptive Behavior in Children and Adolescents with Autism Spectrum Disorder: Effects on Sleep Parameters as Measured by the CSHQ. *Biomedicines*. Jul 13 2022;10(7)doi:10.3390/biomedicines10071685
- 10. Aran A, Cayam Rand D. Cannabinoid treatment for the symptoms of autism spectrum disorder. *Expert Opin Emerg Drugs*. Mar 2024;29(1):65-79. doi:10.1080/14728214.2024.2306290
- 11. Guerrero-Alba R, Barragan-Iglesias P, Gonzalez-Hernandez A, et al. Some Prospective Alternatives for Treating Pain: The Endocannabinoid System and Its Putative Receptors GPR18 and GPR55. *Front Pharmacol*. 2018;9:1496. doi:10.3389/fphar.2018.01496
- 12. Melancia F, Schiavi S, Servadio M, et al. Sex-specific autistic endophenotypes induced by prenatal exposure to valproic acid involve anandamide signalling. *Br J Pharmacol*. Sep 2018;175(18):3699-3712. doi:10.1111/bph.14435
- 13. Zamberletti E, Gabaglio M, Parolaro D. The Endocannabinoid System and Autism Spectrum Disorders: Insights from Animal Models. *Int J Mol Sci.* Sep 07 2017;18(9)doi:10.3390/ijms18091916

- 14. Wang W, Cox BM, Jia Y, et al. Treating a novel plasticity defect rescues episodic memory in Fragile X model mice. *Mol Psychiatry*. Aug 2018;23(8):1798-1806. doi:10.1038/mp.2017.221
- 15. Hosie S, Malone DT, Liu S, et al. Altered Amygdala Excitation and CB1 Receptor Modulation of Aggressive Behavior in the Neuroligin-3(R451C) Mouse Model of Autism. *Front Cell Neurosci*. 2018;12:234. doi:10.3389/fncel.2018.00234
- 16. Zou M, Liu Y, Xie S, et al. Alterations of the endocannabinoid system and its therapeutic potential in autism spectrum disorder. *Open Biol*. Feb 2021;11(2):200306. doi:10.1098/rsob.200306
- 17. Poleg S, Kourieh E, Ruban A, et al. Behavioral aspects and neurobiological properties underlying medical cannabis treatment in Shank3 mouse model of autism spectrum disorder. *Transl Psychiatry*. Oct 13 2021;11(1):524. doi:10.1038/s41398-021-01612-3
- 18. Karhson DS, Krasinska KM, Dallaire JA, et al. Plasma anandamide concentrations are lower in children with autism spectrum disorder. *Mol Autism*. 2018;9:18. doi:10.1186/s13229-018-0203-y
- 19. Aran A, Eylon M, Harel M, et al. Lower circulating endocannabinoid levels in children with autism spectrum disorder. *Mol Autism*. 2019;10:2. doi:10.1186/s13229-019-0256-6
- 20. Szkudlarek HJ, Desai SJ, Renard J, et al. Delta-9-Tetrahydrocannabinol and Cannabidiol produce dissociable effects on prefrontal cortical executive function and regulation of affective behaviors. *Neuropsychopharmacology*. Mar 2019;44(4):817-825. doi:10.1038/s41386-018-0282-7
- 21. Campos AC, Fogaca MV, Scarante FF, et al. Plastic and Neuroprotective Mechanisms Involved in the Therapeutic Effects of Cannabidiol in Psychiatric Disorders. *Front Pharmacol*. 2017;8:269. doi:10.3389/fphar.2017.00269
- 22. McGuire P, Robson P, Cubala WJ, et al. Cannabidiol (CBD) as an Adjunctive Therapy in Schizophrenia: A Multicenter Randomized Controlled Trial. *Am J Psychiatry*. Mar 1 2018;175(3):225-231. doi:10.1176/appi.ajp.2017.17030325
- 23. Devinsky O, Cilio MR, Cross H, et al. Cannabidiol: pharmacology and potential therapeutic role in epilepsy and other neuropsychiatric disorders. *Epilepsia*. Jun 2014;55(6):791-802. doi:10.1111/epi.12631
- 24. Iannotti FA, Hill CL, Leo A, et al. Nonpsychotropic plant cannabinoids, cannabidivarin (CBDV) and cannabidiol (CBD), activate and desensitize transient receptor potential vanilloid 1 (TRPV1) channels in vitro: potential for the treatment of neuronal hyperexcitability. *ACS Chem Neurosci*. Nov 19 2014;5(11):1131-41. doi:10.1021/cn5000524
- 25. Cifelli P, Ruffolo G, De Felice E, et al. Phytocannabinoids in Neurological Diseases: Could They Restore a Physiological GABAergic Transmission? *Int J Mol Sci*. Jan 22 2020;21(3)doi:10.3390/ijms21030723
- 26. Atalay S, Jarocka-Karpowicz I, Skrzydlewska E. Antioxidative and Anti-Inflammatory Properties of Cannabidiol. *Antioxidants (Basel)*. Dec 25 2019;9(1)doi:10.3390/antiox9010021
- 27. Ribeiro A, Ferraz-de-Paula V, Pinheiro ML, et al. Cannabidiol, a non-psychotropic plant-derived cannabinoid, decreases inflammation in a murine model of

- acute lung injury: role for the adenosine A(2A) receptor. Eur J Pharmacol. Mar 5 2012;678(1-3):78-85. doi:10.1016/j.ejphar.2011.12.043
- 28. Furgiuele A, Cosentino M, Ferrari M, Marino F. Immunomodulatory Potential of Cannabidiol in Multiple Sclerosis: a Systematic Review. *J Neuroimmune Pharmacol*. Jan 25 2021:1-19. doi:10.1007/s11481-021-09982-7
- 29. Kozela E, Lev N, Kaushansky N, et al. Cannabidiol inhibits pathogenic T cells, decreases spinal microglial activation and ameliorates multiple sclerosis-like disease in C57BL/6 mice. *Br J Pharmacol*. Aug 2011;163(7):1507-19. doi:10.1111/j.1476-5381.2011.01379.x
- 30. Kozela E, Juknat A, Kaushansky N, Rimmerman N, Ben-Nun A, Vogel Z. Cannabinoids decrease the th17 inflammatory autoimmune phenotype. *J Neuroimmune Pharmacol*. Dec 2013;8(5):1265-76. doi:10.1007/s11481-013-9493-1
- 31. Kozela E, Juknat A, Gao F, Kaushansky N, Coppola G, Vogel Z. Pathways and gene networks mediating the regulatory effects of cannabidiol, a nonpsychoactive cannabinoid, in autoimmune T cells. *J Neuroinflammation*. Jun 3 2016;13(1):136. doi:10.1186/s12974-016-0603-x
- 32. Burstein S. Cannabidiol (CBD) and its analogs: a review of their effects on inflammation. *Bioorg Med Chem.* Apr 1 2015;23(7):1377-85. doi:10.1016/j.bmc.2015.01.059
- 33. Mecha M, Feliú A, Iñigo PM, Mestre L, Carrillo-Salinas FJ, Guaza C. Cannabidiol provides long-lasting protection against the deleterious effects of inflammation in a viral model of multiple sclerosis: a role for A2A receptors. *Neurobiol Dis.* Nov 2013;59:141-50. doi:10.1016/j.nbd.2013.06.016
- 34. Kozela E, Pietr M, Juknat A, Rimmerman N, Levy R, Vogel Z. Cannabinoids Delta(9)-tetrahydrocannabinol and cannabidiol differentially inhibit the lipopolysaccharide-activated NF-kappaB and interferon-beta/STAT proinflammatory pathways in BV-2 microglial cells. *J Biol Chem.* Jan 15 2010;285(3):1616-26. doi:10.1074/jbc.M109.069294
- 35. Juknat A, Pietr M, Kozela E, et al. Differential transcriptional profiles mediated by exposure to the cannabinoids cannabidiol and  $\Delta 9$ -tetrahydrocannabinol in BV-2 microglial cells. *Br J Pharmacol*. Apr 2012;165(8):2512-28. doi:10.1111/j.1476-5381.2011.01461.x
- 36. Juknat A, Pietr M, Kozela E, et al. Microarray and pathway analysis reveal distinct mechanisms underlying cannabinoid-mediated modulation of LPS-induced activation of BV-2 microglial cells. *PLoS One*. 2013;8(4):e61462. doi:10.1371/journal.pone.0061462
- 37. Juknat A, Gao F, Coppola G, Vogel Z, Kozela E. miRNA expression profiles and molecular networks in resting and LPS-activated BV-2 microglia-Effect of cannabinoids. *PLoS One*. 2019;14(2):e0212039. doi:10.1371/journal.pone.0212039
- 38. Zengeler KE, Lukens JR. Innate immunity at the crossroads of healthy brain maturation and neurodevelopmental disorders. *Nat Rev Immunol*. Jan 21 2021;doi:10.1038/s41577-020-00487-7
- 39. Morgan JT, Chana G, Pardo CA, et al. Microglial activation and increased microglial density observed in the dorsolateral prefrontal cortex in autism. *Biol Psychiatry*. Aug 15 2010;68(4):368-76. doi:10.1016/j.biopsych.2010.05.024

- 40. Vargas DL, Nascimbene C, Krishnan C, Zimmerman AW, Pardo CA. Neuroglial activation and neuroinflammation in the brain of patients with autism. *Ann Neurol*. Jan 2005;57(1):67-81. doi:10.1002/ana.20315
- 41. Tetreault NA, Hakeem AY, Jiang S, et al. Microglia in the cerebral cortex in autism. *J Autism Dev Disord*. Dec 2012;42(12):2569-84. doi:10.1007/s10803-012-1513-0
- 42. Gupta S, Ellis SE, Ashar FN, et al. Transcriptome analysis reveals dysregulation of innate immune response genes and neuronal activity-dependent genes in autism. *Nat Commun.* Dec 10 2014;5:5748. doi:10.1038/ncomms6748
- 43. Suzuki K, Sugihara G, Ouchi Y, et al. Microglial activation in young adults with autism spectrum disorder. *JAMA Psychiatry*. Jan 2013;70(1):49-58. doi:10.1001/jamapsychiatry.2013.272
- 44. Voineagu I, Wang X, Johnston P, et al. Transcriptomic analysis of autistic brain reveals convergent molecular pathology. *Nature*. May 25 2011;474(7351):380-4. doi:10.1038/nature10110
- 45. Goines PE, Ashwood P. Cytokine dysregulation in autism spectrum disorders (ASD): possible role of the environment. *Neurotoxicol Teratol*. Mar-Apr 2013;36:67-81. doi:10.1016/j.ntt.2012.07.006
- 46. Onore C, Careaga M, Ashwood P. The role of immune dysfunction in the pathophysiology of autism. *Brain Behav Immun*. Mar 2012;26(3):383-92. doi:10.1016/j.bbi.2011.08.007
- 47. Griffiths KK, Levy RJ. Evidence of Mitochondrial Dysfunction in Autism: Biochemical Links, Genetic-Based Associations, and Non-Energy-Related Mechanisms. *Oxidative Medicine and Cellular Longevity*. 2017/05/29 2017;2017:4314025. doi:10.1155/2017/4314025
- 48. Singh K, Singh IN, Diggins E, et al. Developmental regression and mitochondrial function in children with autism. *Ann Clin Transl Neurol*. May 2020;7(5):683-694. doi:10.1002/acn3.51034
- 49. Jyonouchi H, Geng L, Rose S, Bennuri SC, Frye RE. Variations in Mitochondrial Respiration Differ in IL-1B/IL-10 Ratio Based Subgroups in Autism Spectrum Disorders. *Front Psychiatry*. 2019;10:71. doi:10.3389/fpsyt.2019.00071
- 50. Aran A, Harel M, Cassuto H, et al. Cannabinoid treatment for autism: a proof-of-concept randomized trial. *Mol Autism*. Feb 3 2021;12(1):6. doi:10.1186/s13229-021-00420-2
- 51. clinicaltrials g. <a href="https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist="https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&cntry=&state=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=CBD&term=CBD&term=&city=&city=&dist==."https://clinicaltrials.gov/ct2/results?cond=ASD&term=&city=
- 52. Raz N, Eyal AM, Davidson EM. Optimal Treatment with Cannabis Extracts Formulations Is Gained via Knowledge of Their Terpene Content and via Enrichment with Specifically Selected Monoterpenes and Monoterpenoids. *Molecules*. Oct 15 2022;27(20)doi:10.3390/molecules27206920
- 53. Staben J, Koch M, Reid K, et al. Cannabidiol and cannabis-inspired terpene blends have acute prosocial effects in the BTBR mouse model of autism spectrum disorder. *Front Neurosci.* 2023;17:1185737. doi:10.3389/fnins.2023.1185737

- 54. Raz N, Eyal AM, Zeitouni DB, et al. Selected cannabis terpenes synergize with THC to produce increased CB1 receptor activation. *Biochem Pharmacol*. Jun 2023;212:115548. doi:10.1016/j.bcp.2023.115548
- 55. Câmara JS, Perestrelo R, Ferreira R, Berenguer CV, Pereira JAM, Castilho PC. Plant-Derived Terpenoids: A Plethora of Bioactive Compounds with Several Health Functions and Industrial Applications-A Comprehensive Overview. *Molecules*. Aug 15 2024;29(16)doi:10.3390/molecules29163861
- 56. Rava A, Buzzelli V, Feo A, et al. Role of peroxisome proliferator-activated receptors  $\alpha$  and  $\gamma$  in mediating the beneficial effects of  $\beta$ -caryophyllene in a rat model of fragile X syndrome. *Prog Neuropsychopharmacol Biol Psychiatry*. Jan 10 2025;136:111234. doi:10.1016/j.pnpbp.2024.111234
- 57. Alayoubi M, Rodrigues A, Wu C, et al. Elucidating interplay between myrcene and cannabinoid receptor 1 receptors to produce antinociception in mouse models of neuropathic pain. *Pain*. Mar 18 2025;doi:10.1097/j.pain.0000000000003558
- 58. McCracken JT, McGough J, Shah B, et al. Risperidone in children with autism and serious behavioral problems. *The New England journal of medicine*. Aug 1 2002;347(5):314-21. doi:10.1056/NEJMoa013171
- 59. Shea S, Turgay A, Carroll A, et al. Risperidone in the treatment of disruptive behavioral symptoms in children with autistic and other pervasive developmental disorders. *Pediatrics*. Nov 2004;114(5):e634-41. doi:10.1542/peds.2003-0264-F
- 60. Levine SZ, Kodesh A, Goldberg Y, et al. Initial severity and efficacy of risperidone in autism: Results from the RUPP trial. *European psychiatry : the journal of the Association of European Psychiatrists*. Feb 2016;32:16-20. doi:10.1016/j.eurpsy.2015.11.004
- 61. Adler BA, Wink LK, Early M, et al. Drug-refractory aggression, self-injurious behavior, and severe tantrums in autism spectrum disorders: a chart review study. *Autism : the international journal of research and practice*. Jan 2015;19(1):102-6. doi:10.1177/1362361314524641
- 62. Taylor L, Gidal B, Blakey G, Tayo B, Morrison G. A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Dose, and Food Effect Trial of the Safety, Tolerability and Pharmacokinetics of Highly Purified Cannabidiol in Healthy Subjects. *CNS Drugs*. Nov 2018;32(11):1053-1067. doi:10.1007/s40263-018-0578-5
- 63. Voinsky I, Zoabl Y, Shomron N, et al. Blood

RNA sequencing confirms upregulated BATF2 and FCGR1A expression in children

with autism spectrum disorder. <a href="https://www.researchsquare.com/article/rs-1113898/v1">https://www.researchsquare.com/article/rs-1113898/v1</a>; 2021.

- 64. Siani-Rose M, Cox S, Goldstein B, Abrams D, Taylor M, Kurek I. Cannabis-Responsive Biomarkers: A Pharmacometabolomics-Based Application to Evaluate the Impact of Medical Cannabis Treatment on Children with Autism Spectrum Disorder. *Cannabis Cannabinoid Res.* Dec 6 2021;doi:10.1089/can.2021.0129
- 65. Iglesias-Vázquez L, Van Ginkel Riba G, Arija V, Canals J. Composition of Gut Microbiota in Children with Autism Spectrum Disorder: A Systematic Review and Meta-Analysis. *Nutrients*. Mar 17 2020;12(3)doi:10.3390/nu12030792

- 66. Sharon G, Cruz NJ, Kang DW, et al. Human Gut Microbiota from Autism Spectrum Disorder Promote Behavioral Symptoms in Mice. *Cell*. May 30 2019;177(6):1600-1618.e17. doi:10.1016/j.cell.2019.05.004
- 67. Ding X, Xu Y, Zhang X, et al. Gut microbiota changes in patients with autism spectrum disorders. *J Psychiatr Res*. Oct 2020;129:149-159. doi:10.1016/j.jpsychires.2020.06.032
- 68. Schopler E, Reichler RJ, DeVellis RF, Daly K. Toward objective classification of childhood autism: Childhood Autism Rating Scale (CARS). *Journal of autism and developmental disorders*. Mar 1980;10(1):91-103.
- 69. Nader AM, Courchesne V, Dawson M, Soulières I. Does WISC-IV Underestimate the Intelligence of Autistic Children? *J Autism Dev Disord*. May 2016;46(5):1582-9. doi:10.1007/s10803-014-2270-z
- 70. Dawson M, Soulières I, Gernsbacher MA, Mottron L. The level and nature of autistic intelligence. *Psychol Sci.* Aug 2007;18(8):657-62. doi:10.1111/j.1467-9280.2007.01954.x
- 71. Courchesne V, Meilleur AA, Poulin-Lord MP, Dawson M, Soulières I. Autistic children at risk of being underestimated: school-based pilot study of a strength-informed assessment. *Mol Autism.* 2015;6:12. doi:10.1186/s13229-015-0006-3
- 72. Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. *American journal of mental deficiency*. Mar 1985;89(5):485-91.
- 73. Aman M. Aberrant behaviour checklist—community. East Aurora, NY: Slosson Educational Publications; 1994.
- 74. Fung LK, Mahajan R, Nozzolillo A, et al. Pharmacologic Treatment of Severe Irritability and Problem Behaviors in Autism: A Systematic Review and Meta-analysis. *Pediatrics*. Feb 2016;137 Suppl 2:S124-35. doi:10.1542/peds.2015-2851K
- 75. Taylor J, Watkins C, Kaplin A. Kleine-Levin syndrome: a disease in its own right? *Nat Clin Pract Neurol*. Oct 2008;4(10):534-5. doi:ncpneuro0900 [pii]

### 10.1038/ncpneuro0900 [doi]

- 76. Constantino JN, Gruber CP. The Social Responsiveness Scale (SRS) (Manual). Los Angeles: Western Psychological Services. 2005;
- 77. Ben-Sasson A, Lamash L, Gal E. To enforce or not to enforce? The use of collaborative interfaces to promote social skills in children with high functioning autism spectrum disorder. *Autism: the international journal of research and practice*. Sep 2013;17(5):608-22. doi:10.1177/1362361312451526
- 78. Aman MG, Findling RL, Hardan AY, et al. Safety and Efficacy of Memantine in Children with Autism: Randomized, Placebo-Controlled Study and Open-Label Extension. *Journal of child and adolescent psychopharmacology*. Mar 15 2016;doi:10.1089/cap.2015.0146
- 79. Freitag CM, Jensen K, Elsuni L, et al. Group-based cognitive behavioural psychotherapy for children and adolescents with ASD: the randomized, multicentre, controlled SOSTA net trial. *Journal of child psychology and psychiatry, and allied disciplines*. May 2016;57(5):596-605. doi:10.1111/jcpp.12509

- 80. Minshawi NF, Wink LK, Shaffer R, et al. A randomized, placebo-controlled trial of D-cycloserine for the enhancement of social skills training in autism spectrum disorders. *Molecular autism*. 2016;7:2. doi:10.1186/s13229-015-0062-8
- 81. Hendren RL, James SJ, Widjaja F, Lawton B, Rosenblatt A, Bent S. Randomized, Placebo-Controlled Trial of Methyl B12 for Children with Autism. *Journal of child and adolescent psychopharmacology*. Feb 18 2016;doi:10.1089/cap.2015.0159
- 82. Fujioka T, Inohara K, Okamoto Y, et al. Gazefinder as a clinical supplementary tool for discriminating between autism spectrum disorder and typical development in male adolescents and adults. *Molecular autism*. 2016;7:19. doi:10.1186/s13229-016-0083-y
- 83. Bone D, Bishop S, Black MP, Goodwin MS, Lord C, Narayanan SS. Use of machine learning to improve autism screening and diagnostic instruments: effectiveness, efficiency, and multi-instrument fusion. *Journal of child psychology and psychiatry, and allied disciplines*. Apr 19 2016;doi:10.1111/jcpp.12559
- 84. Guy W. ECDEU Assessment Manual for Psychopharmacology: Publication ADM 76-338. Washington, DC: US Dept of Health, Education, and Welfare. 1976:218-222.
- 85. King BH, Hollander E, Sikich L, et al. Lack of efficacy of citalopram in children with autism spectrum disorders and high levels of repetitive behavior: citalopram ineffective in children with autism. *Archives of general psychiatry*. Jun 2009;66(6):583-90. doi:10.1001/archgenpsychiatry.2009.30
- 86. Bearss K, Johnson C, Smith T, et al. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. *Jama*. Apr 21 2015;313(15):1524-33. doi:10.1001/jama.2015.3150
- 87. Mazurek MO, Carlson C, Baker-Ericzén M, Butter E, Norris M, Kanne S. Construct Validity of the Autism Impact Measure (AIM). *J Autism Dev Disord*. Jul 2020;50(7):2307-2319. doi:10.1007/s10803-018-3462-8
- 88. Silkey M, Durán-Pacheco G, Johnson M, et al. The Autism Impact Measure (AIM): Meaningful Change Thresholds and Core Symptom Changes Over One Year from an Online Survey in the U.S. *J Autism Dev Disord*. Sep 2023;53(9):3422-3434. doi:10.1007/s10803-022-05635-7
- 89. Wakschlag LS, Briggs-Gowan MJ, Choi SW, et al. Advancing a multidimensional, developmental spectrum approach to preschool disruptive behavior. *J Am Acad Child Adolesc Psychiatry*. Jan 2014;53(1):82-96.e3. doi:10.1016/j.jaac.2013.10.011
- 90. Mazefsky CA, Yu L, White SW, Siegel M, Pilkonis PA. The emotion dysregulation inventory: Psychometric properties and item response theory calibration in an autism spectrum disorder sample. *Autism Res.* Jun 2018;11(6):928-941. doi:10.1002/aur.1947
- 91. Aita SL, Moncrief GG, Greene J, et al. Univariate and Multivariate Base Rates of Score Elevations, Reliable Change, and Inter-Rater Discrepancies in the BRIEF-A Standardization Samples. *Assessment*. Mar 2023;30(2):390-401. doi:10.1177/10731911211055673
- 92. Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. *Sleep*. Dec 15 2000;23(8):1043-51.

- 93. Eapen V, Crnčec R, Walter A, Tay KP. Conceptualisation and development of a quality of life measure for parents of children with autism spectrum disorder. *Autism Res Treat*. 2014;2014:160783. doi:10.1155/2014/160783
- 94. Margolis KG, Buie TM, Turner JB, et al. Development of a Brief Parent-Report Screen for Common Gastrointestinal Disorders in Autism Spectrum Disorder. *J Autism Dev Disord*. Jan 2019;49(1):349-362. doi:10.1007/s10803-018-3767-7
- 95. Zimmerman AW, Singh K, Connors SL, et al. Randomized controlled trial of sulforaphane and metabolite discovery in children with Autism Spectrum Disorder. *Mol Autism*. May 25 2021;12(1):38. doi:10.1186/s13229-021-00447-5
- 96. Fallah MS, Shaikh MR, Neupane B, Rusiecki D, Bennett TA, Beyene J. Atypical Antipsychotics for Irritability in Pediatric Autism: A Systematic Review and Network Meta-Analysis. *J Child Adolesc Psychopharmacol*. Apr 2019;29(3):168-180. doi:10.1089/cap.2018.0115
- 97. Gaston TE, Ampah SB, Martina Bebin E, et al. Long-term safety and efficacy of highly purified cannabidiol for treatment refractory epilepsy. *Epilepsy Behav*. Apr 2021;117:107862. doi:10.1016/j.yebeh.2021.107862
- 98. Thiele EA, Bebin EM, Filloux F, et al. Long-term cannabidiol treatment for seizures in patients with tuberous sclerosis complex: An open-label extension trial. *Epilepsia*. Dec 27 2021;doi:10.1111/epi.17150
- 99. Patel AD, Mazurkiewicz-Bełdzińska M, Chin RF, et al. Long-term safety and efficacy of add-on cannabidiol in patients with Lennox-Gastaut syndrome: Results of a long-term open-label extension trial. *Epilepsia*. Sep 2021;62(9):2228-2239. doi:10.1111/epi.17000
- 100. Scheffer IE, Halford JJ, Miller I, et al. Add-on cannabidiol in patients with Dravet syndrome: Results of a long-term open-label extension trial. *Epilepsia*. Oct 2021;62(10):2505-2517. doi:10.1111/epi.17036
- 101. Devinsky O, Patel AD, Cross JH, et al. Effect of Cannabidiol on Drop Seizures in the Lennox-Gastaut Syndrome. *N Engl J Med*. May 17 2018;378(20):1888-1897. doi:10.1056/NEJMoa1714631
- 102. Silva EADJ, Medeiros WMB, Santos J, et al. Evaluation of the efficacy and safety of cannabidiol-rich cannabis extract in children with autism spectrum disorder: randomized, double-blind and controlled placebo clinical trial. *Trends Psychiatry Psychother*. May 26 2022;44doi:10.47626/2237-6089-2021-0396